

# Statistical Analysis Plan

| Protocol No | GPL/CT/2014/018/III (Study No. GSP 301-303) |
|---|---|
| Protocol Title | A Double-Blind, Randomized, Parallel-Group Study to Evaluate Long-<br>Term Safety, Tolerability, and Efficacy of a Fixed Dose Combination GSP<br>301 Nasal Spray Compared with Two Placebo Nasal Spray Formulations<br>in Subjects (Aged 12 Years and Older) with Perennial Allergic Rhinitis<br>(PAR) |
| Protocol version | Version 2.0 |
| Sponsor | Glenmark Specialty S.A. Avenue Léopold-Robert 37 2300 La Chaux-de-Fonds Switzerland |

# **Document Version History**

| Version<br>Number | Version Date | Description of change |
|-------------------|--------------|-----------------------|
| 1.0 | 04-Apr-2017 | New Document |



# **Review and Approval Page**

The signatures on this page indicate review and approval of Statistical Analysis Plan.

| I have reviewed the above-mentioned version of Statistical Analysis Plan and confirm it to be complete and accurate. | | |
|---|---|---|
| Prepared by: | | |
| Senior Biostatistician | Signature: | OH/APR/2017 Date (DD/MMM/YYYY): |
| Approval | | |
| Director of Statistical Science | | |
| | Signature: | Date (DD/MMM/YYYY): 05/ Apr.4/2017 |



Protocol Number: GPL/CT/2014/018/III (Study No. GSP 301-303) SAP Version Number:

Version 1.0 04-

SAP Version Date: 04-Apr-2017

## **Abbreviations and Specialist Terms**

| ADaM | Analysis Data Model |
|---|---|
| AE | Adverse Event |
| AM | Morning |
| AESI | Adverse Events of Special Interest |
| ANCOVA | Analysis of Covariance |
| AR | Allergic rhinitis |
| BDRM | Blinded Data Review Meeting |
| BID | Twice Daily Dosing |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| CS | Clinically Significant |
| CSR | Clinical study report |
| ECG | Electrocardiogram |
| ENT | Ears, nose, and throat |
| °F | Degrees Fahrenheit |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration (of the United States) |
| FDC | Fixed dose combination |
| GSP 301 NS | Fixed Dose Combination of olopatadine hydrochloride and mometasone |
| | furoate nasal spray |
| iTNSS | Instantaneous Total Nasal Symptom Score |
| ICF | Informed consent form |
| ICH | International Conference on Harmonisation |
| ITT | Intent To Treat |
| IP | Investigational product |
| LOCF | Last Observation Carried Forward |
| LSM | Least squares mean |
| μg | Microgram |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed Model Repeated Measures |
| NCS | Not Clinically Significant |
| NS | Nasal Spray |
| PAR | Perennial Allergic Rhinitis |
| PK | Pharmacokinetic |
| PNSS | Physician Assessed Nasal Symptom Score |
| PPS | Per Protocol Set |
| PT | Preferred Term |
| RCAT | Rhinitis Control Assessment Test |



Protocol Number: GPL/CT/2014/018/III (Study No. GSP 301-303) SAP Version Number: Version 1.0

SAP Version Date:

04-Apr-2017

| RQLQ(S) | Rhinoconjuntivitis Quality of Life Questionnaire Standardized Activities |
|---|---|
| rTNSS | Reflective Total Nasal Symptom Score |
| QD | Once Daily Dosing |
| SAEs | Serious Adverse Events |
| SAP | Statistical Analysis Plan |
| SAR | Seasonal Allergic Rhinitis |
| SAS | Statistical Analysis System |
| SAS | Safety Analysis Set |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| SPT | Skin Prick Test |
| TEAE | Treatment-emergent Adverse Event |
| TNSS | Total Nasal Symptom Score |




04-Apr-2017

| | Changes to the Protocol Defined Statistical Analysis Plan | |
|---|---|---|
| | Introduction | |
| | Objectives | |
| 3.1 | Primary Objective | . 8 |
| 3.2 | Secondary Objective(s) | . 8 |
| 4.0 | Study Endpoints | . 8 |
| 4.1 | Primary Endpoints | . 8 |
| 4.2 | Secondary Endpoints | . 8 |
| | Study Design | |
| | Statistical Hypotheses | |
| | Randomization and Blinding | |
| | Sample Size Determination | |
| | Planned Analyses | |
| | Interim Analyses | |
| | Final Analyses | |
| | Analysis Sets | |
| | Efficacy Assessments and Derivation of Endpoints | |
| | Subject-Reported Nasal Symptoms | |
| | Rhinoconjunctivitis Quality-Of-Life Questionnaire - Standardized Activities (RQLQ(S)) | |
| | Physician Assessed Nasal Symptom Score (PNSS) | |
| | Rhinitis Control Assessment Test (RCAT) | |
| | Statistical Analysis Methods | |
| | Study Population Analyses | |
| 12.1.1 | Overview of Planned Analyses | 16 |
| 12.1.2 | Supplementary Information for Study Population Tables and Listings | 17 |
| 12.1.2. | 1 Subject Disposition | 17 |
| 12.1.2.2 | | |
| | 3 Medical History | |
| | 4 Extent of Exposure | |
| | 5 Concomitant Medications | |
| 12.2 | Safety Analyses | |
| 12.2.1 | the state of the s | |
| | Adverse Events | |
| | Adverse Events of Special Interest (AESI) | |
| | Laboratory Data | |
| | Pregnancy Test | |
| | Vital Signs | |
| 12.2.7 | | |
| 12.2.8 | <b>)</b> | |
| 12.2.9 | | |
| 12.2.10 | Rescue Medication | 24 |




| 12.3 | Efficacy Analyses of Efficacy Endpoints | 25 |
|---|---|---|
| | Overview of Efficacy Analysis of the Efficacy Endpoints (rTNSS, iTNSS, F | |
| | the first 6, 30, and 52 weeks of treatment) | 25 |
| 12.3.2 | Analysis Method of the Efficacy Endpoints (rTNSS, iTNSS, RQLQ(S)): Mi | xed Model |
| | Repeated Measures Approach | 26 |
| 12.3.6 | Examination of Subgroups | 29 |
| 12.4 | Efficacy Analyses of Other Efficacy Endpoints | 29 |
| 12.4.1 | Overview of Analysis of the Other Efficacy Endpoints | 29 |
| 12.4.2 | Analysis of Change from Baseline in Other Efficacy Endpoints | 32 |
| Append | dix 1 | 35 |
| Refere | nce: | 148 |
| Append | dix 2 | 149 |




#### 1.0 Changes to the Protocol Defined Statistical Analysis Plan

- The protocol states that the efficacy analysis will be conducted using an analysis of covariance (ANCOVA) model (adjusting for study treatment group, site and baseline).
   The efficacy analysis will now be analyzed using a mixed models repeated measures (MMRM) model. This will be more applicable to the design of the study, and assesses missing data using the Missing at Random (MAR) assumption. More detail is in Section 12.3.
- The protocol states that 'A multiple, imputation-based approach where complete data sets are drawn will be used for handling missing data in the efficacy analysis.' Because assessing efficacy is a secondary objective of the study, the sentence has been modified to state 'A multiple, imputation-based approach may be considered for handling missing data for AM reflective Total Nasal Symptom Score (rTNSS) and AM instantaneous Total Nasal Symptom Score (iTNSS) upon review of amount of missing data observed'. More details in Section 12.3.
- The protocol states that the computer-generated randomization scheme will be reviewed and approved by an independent statistician and the randomization will be stratified by site. This was inaccurately stated. The computer-generated randomization scheme will be reviewed and approved by a statistician and the randomization will not be stratified by site. More detail is in Section 7.0.
- The protocol has defined the Full Analysis Set (FAS) as 'The FAS will consist of all subjects who are randomized and received at least 1 dose of Investigational Product (IP) and have at least 1 post-baseline efficacy assessment.' To add more clarity the definition of the FAS is 'The FAS will consist of all subjects who are randomized and received at least 1 dose of IP and have at least 1 post-baseline AM rTNSS assessment.

#### 2.0 Introduction

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol GPL/CT/2014/018/III Version 2.0 (Study No. GSP 301-303) dated 31-Aug-2016. The SAP provides details of the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

 Final Clinical Study Protocol GPL/CT/2014/018/III Version 2.0 (Study No. GSP 301-303) dated 31-Aug-2016

|--------------------------|--------------|---------------|
|--------------------------|--------------|---------------|



Protocol Number: GPL/CT/2014/018/III SAP Version Number: Version 1.0


(Study No. GSP 301-303)

04-Apr-2017

GSP 301-303 final CRF dated 19-May-2016

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a subject in this study.

#### 3.0 Objectives

#### 3.1 Primary Objective

 To compare the long-term safety and tolerability of GSP 301 NS with 2 GSP 301 placebo NS formulations over 52 weeks of study treatment

#### 3.2 Secondary Objective(s)

 To evaluate the long-term efficacy of GSP 301 NS compared with GSP 301 placebo in subjects with Perennial Allergic Rhinitis (PAR).

#### 4.0 Study Endpoints

#### 4.1 Primary Endpoints

- Proportion of subjects with treatment-emergent adverse events (TEAEs).
- Proportion of subjects with treatment-related TEAEs.
- Incidence, type, and severity of the TEAEs after 30 weeks of study treatment.
- Incidence, type, and severity of the TEAEs after 52 weeks of study treatment.
- Clinical laboratory assessments (hematology, serum biochemistry, and urinalysis) at baseline, Week 30, and Week 52.
- Vital signs, physical examinations (PE), and focused ears, nose, and throat (ENT) and eye examinations at baseline, Week 30, and Week 52.

#### 4.2 Secondary Endpoints

#### **Efficacy Endpoints:**

- Change from baseline in the average AM subject-reported rTNSS over the first 6, 30, and 52 weeks of treatment.
- Change from baseline in the average AM subject-reported instantaneous Total Nasal Symptom Score (iTNSS) over the first 6, 30, and 52 weeks of treatment.
- Change from baseline in the overall Rhinoconjunctivitis Quality of Life Questionnaire - Standardized Activities (RQLQ(S)) score at Weeks 6, 30, and 52 for the Full Analysis Set (FAS).




Version 1.0


#### Other Efficacy Endpoints:

#### **Nasal symptoms:**

- Change from baseline in the average AM subject-reported reflective individual nasal symptoms over the first 6, 30, and 52 weeks of treatment.
- Change from baseline in the average AM subject-reported instantaneous individual nasal symptoms over the first 6, 30, and 52 weeks of treatment.
- Change in the average AM subject-reported rTNSS and iTNSS from baseline to the end of each treatment week.
- Change in the average AM subject-reported reflective individual nasal symptoms from baseline to the end of each treatment week.
- Change in the average AM subject-reported instantaneous individual nasal symptoms from baseline to the end of each treatment week.

Physician assessed Nasal Symptom Score (PNSS), Rhinoconjunctivitis Quality of Life Questionnaire – Standardized Activities (RQLQ(S)), and Rhinitis Control Assessment Test (RCAT):

- Change from baseline in PNSS and physician assessed individual nasal symptoms at Weeks 6, 30, and 52.
- Change from baseline in individual domains of the RQLQ(S) at Weeks 6, 30, and 52 for the FAS.
- Change from baseline in overall RQLQ(S) score and individual domains of the RQLQ(S) at Weeks 6, 30, and 52 for the RQLQ(S) Analysis Set.
- Change from baseline in the RCAT at Weeks 6, 30, and 52.
- Change from baseline in individual domains of the RCAT at Weeks 6, 30, and 52.

#### 5.0 Study Design

This is a multi-center, double-blind, randomized, parallel-group, 52-week study conducted in subjects with PAR. The subjects will be randomized to the following 3 treatment groups in a ratio of 4:1:1:

- GSP 301 NS (665 μg olopatadine hydrochloride/25 μg mometasone furoate)
   administered as
- GSP 301 placebo NS pH administered as
- GSP 301 placebo NS pH
   administered as

This study consists of 12 visits to the study site (Figure 1). After the initial Screening Visit (Visit 1), subjects who meet all study selection criteria will undergo a single-blind, placebo, run-in period for 7 to 10 days. Following the completion of the run-in period, eligible subjects who meet the randomization criteria will be enrolled and randomized to 1 of the 3 treatment




groups. Randomized subjects will undergo a 52-week treatment period to assess the efficacy and safety of the assigned treatment.

Figure 1: Study Design Schematic



The Screening Visit (Visit 1) will occur 7 to 10 days before the Randomization Visit (Visit 2). The purposes of the Screening Visit (Visit 1) are to obtain informed consent, establish protocol eligibility, and enter eligible subjects into the placebo run-in period. Informed consent will be obtained after the study has been fully explained to each subject and before the conduct of any screening procedures or assessments. The Screening Disposition case report form/electronic case report form (CRF/eCRF) page must be completed to indicate whether the subject is eligible to participate in the study and to provide reasons for screen failure, if applicable. Eligible subjects will be given an AR Assessment Diary to record AR symptoms (morning [AM] rTNSS and iTNSS) during the 7 to 10 day run-in period.

After screening, all eligible subjects will participate in a single-blind, placebo (GSP 301 placebo NS pH run-in period. This is to familiarize the subjects to study procedures (such as study drug administration and symptom assessments) and to identify any potentially non-compliant subjects. The form of single-blind study medication will be taken immediately after completing the diary. The form of the single-blind study medication will be taken approximately 12 hours after the Subjects must meet the key randomization criteria required for the run-in period (m n mum AM subject-reported rTNSS, AM subject-reported reflective nasal congestion score, adequate AR Assessment Diary compliance, and compliance with avoiding prohibited concomitant medications) to continue in the study.

The treatment period consists of 52 weeks. During this time, subjects will continue to assess their symptoms and complete the AR Assessment Diary every morning. The dose of double-blind study medication will be taken immediately after completing the diary. The dose of the single-blind study medication will be taken

The last dose of study medication should be the Final Visit/Discontinuation Visit (Visit 12).




No scheduled post-treatment follow-up visit is planned for this study. However, subjects will be followed up if there is any ongoing AE or for any other reason as per the Investigator's and Sponsor's discretion.

A telephone follow-up will be carried out for this study for any reason as per the Investigator's judgment. If needed, additional unscheduled visits may be conducted to ensure subject safety or to perform other study-related procedures at the discretion of the Investigator or the Sponsor.

No extension phase is planned for this study.

#### 6.0 Statistical Hypotheses

N/A.

#### 7.0 Randomization and Blinding

Subjects will be assigned to 1 of the 3 treatment groups in a 4:1:1 ratio based on a computer-generated randomization scheme that will be reviewed and approved by a statistician.

This study is designed as a double-blind study. The blinding will be maintained by packaging the active products and placebo in identical bottles and outer cartons. Additionally, an unblinded qualified person who is not associated with the study team, will facilitate the randomization process to ensure that the double-blind design of the study is maintained.

#### 8.0 Sample Size Determination

The sample size of 600 subjects for this study (400 subjects on GSP 301 NS and 100 subjects in each of the 2 placebo groups) is based on the ICH E1 Guideline (ICH E1) and the FDA Guidance on Allergic Rhinitis<sup>1</sup> which requires treatment of at least 300 subjects for 6 months and 100 subjects for 1 year. Based on an estimated attrition rate of 25% after 6 months and 50% after 52 weeks, 400 subjects in the GSP 301 NS treatment group are considered sufficient to meet the above requirements.

#### 9.0 Planned Analyses

#### 9.1 Interim Analyses

There is no interim analysis planned in this study.

#### 9.2 Final Analyses

All planned analyses will be carried out once the clinical database lock (DBL) has taken place. Once DBL has been achieved, unblinding will occur and the analyses will be performed.




10.0 Analysis Sets

#### Full Analysis Set (FAS)

The FAS will consist of all subjects who are randomized and received at least 1 dose of IP and have at least 1 post-baseline AM rTNSS assessment. This will be the primary analysis set for efficacy analyses.

#### Per Protocol Set (PPS)

The Per Protocol Set (PPS) will consist of the subset of the FAS who do not meet criteria for PPS exclusion. These criteria are to capture relevant non-adherence to the protocol (defined as a 'major deviation', especially those that affect interpretation of the AM rTNSS endpoint). The PPS will be a secondary analysis set for the efficacy analysis (except for RQLQ(S)). The PPS will be used to assess the robustness of the results from the statistical tests based on the FAS.

Major deviations will lead to the exclusion of a subject from the PPS. Major protocol deviations will be identified during the Blinded Data Review Meeting (BDRM) before database lock.

Major protocol deviations may include:

- Subjects who had their blinded randomization code broken.
- Subjects with overall treatment compliance <75% or >125%.
- Subjects who used prohibited medications (prior and/or concomitant) that may have significant influence on efficacy.
- Subjects who did not satisfy the inclusion/exclusion that may have significant influence on efficacy.
- Subjects not treated with the treatment assigned at randomization, but wrongly treated in another treatment group.

#### Safety Analysis Set (SAS)

The Safety Analysis Set (SAS) will consist of all subjects who took at least 1 dose of study medication following randomization and will be used for all safety analyses.

#### RQLQ(S) Analysis Set

The RQLQ(S) Analysis Set will consist of all English-speaking subjects ≥18 years old with impaired QOL at baseline as defined by a RQLQ(S) score at the Randomization Visit (Visit 2) of 3.0 or greater.




#### 11.0 Efficacy Assessments and Derivation of Endpoints

#### 11.1 Subject-Reported Nasal Symptoms

An efficacy measure in this study is the subject-reported Total Nasal Symptom Score (TNSS). The TNSS is defined as the sum of the subject-reported symptom scores for 4 nasal symptoms: rhinorrhea (runny nose), nasal congestion, nasal itching, and sneezing. The subject will assess and report his/her nasal symptoms in the morning (AM assessment) on each day of the placebo run-in and double-blind treatment periods prior to administering the study treatment. If a nasal symptom score is missing then the TNSS will be set to missing.

The subject will be asked to assess both reflective (i.e., an evaluation of symptom severity over the past 24 hours prior to the recording of the score) and instantaneous (i.e., an evaluation of the symptom severity just before taking study medication nasal symptoms. Each of the following symptoms will be assessed.

Each of the following symptoms will be assessed.

| Nasal Symptoms | |
|------------------------------------------------|-------------|
| 1. Nasal Congestion 2. Rhinorrhea (Runny Nose) | |
| 3. Nasal Itching | 4. Sneezing |

Each of the above symptoms will be rated on a 4-point scale as follows:

| | Grade | Description |
|---|---|---|
| 0 | Absent | No Sign/Symptoms evident |
| 1 | Mild | Sign/Symptoms clearly present but minimal awareness; easily |
| | | tolerated |
| 2 | Moderate | Definite awareness of sign/symptoms which is bothersome but |
| | | tolerable |
| 3 | Severe | Sign/symptoms is hard to tolerate; causes interference with activities of |
| | | daily living and or sleeping |

#### **Derivation Method and Baseline**

#### Mixed Model Repeated Measures (MMRM) Approach

Change from baseline in average AM rTNSS to the end of each treatment week will be derived as the average of post-baseline AM rTNSS scores by week (i.e average AM rTNSS score for Week 1 is calculated as the mean rTNSS score in Week 1), where baseline is defined as the average of the last 4 consecutive AM assessments during the last 4 days of the run-in period from the Day -3 AM assessment to the AM assessment on the day of randomization. At least 2 out of 4 assessments (scores) should be available in order to

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|




calculate the baseline scores for the AM rTNSS. In order to calculate the average of post-baseline AM rTNSS scores by week, at least 2 scores need to be present.

The same derivation method will also be applied to all other nasal symptom efficacy endpoints.

# 11.2 Rhinoconjunctivitis Quality-Of-Life Questionnaire - Standardized Activities (RQLQ(S))

The RQLQ(S) has 28 questions in 7 domains (activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional). Subjects will be asked to recall their experiences during the previous week and to give their responses on a 7-point scale (0=Not troubled to 6=Extremely troubled) for the domains of activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms. The domain "emotional" will utilize a 7-point scale (0=None of the time to 6=All of the time).

RQLQ(S) scores will be summarized by domains. A domain average score is calculated as the sum of the scores in that domain divided by the number of items in that domain; all items in the domain must be valid in order to calculate the corresponding average score. A domain average score will be set to missing if there is a missing item score in that domain.

The overall average RQLQ(S) score is calculated as the sum of the scores in all domains divided by the total number of items in the seven domains; all items in the 7 domains must be valid in order to calculate the corresponding overall average score. If a domain score is missing then the overall average RQLQ(S) score will be set to missing.

Baseline is defined as the RQLQ(S) score at the Randomization Visit (Day 1; Visit 2).

#### 11.3 Physician Assessed Nasal Symptom Score (PNSS)

The Physician-Assessed Total Nasal Symptom Score will be derived from the intensity of the following nasal symptoms associated with AR - rhinorrhea (runny nose), nasal congestion, nasal itching, and sneezing. Physicians will assess severity of the above symptoms for subject-reported nasal symptoms. The PNSS will be based on questioning of the subjects (overall feeling since last visit) and on the ENT examination and other observations by the physician. PNSS is calculated as the sum of the four nasal symptom scores. If a nasal symptom score is missing then the PNSS will be set to missing.

Baseline is defined as the PNSS at the Randomization Visit (Day 1; Visit 2).

#### 11.4 Rhinitis Control Assessment Test (RCAT)

|--------------------------|--------------|----------------|




The Rhinitis Control Assessment Test (RCAT) is a brief, subject-completed tool to evaluate rhinitis symptom control. This questionnaire asks the subject about nasal and other allergy symptoms that are not related to a cold or the flu and the control of these symptoms over the past one week. Responses to the questions are scored by the number next to the response box. The total RCAT score will be calculated by adding individual RCAT item or domain scores. The total RCAT score can range from 6 to 30. If a RCAT item or domain score is missing then the total RCAT score will be set to missing.

Baseline is defined as the RCAT score at the Randomization Visit (Day 1; Visit 2).

#### 12.0 Statistical Analysis Methods

In general, all data will be summarized with descriptive statistics (number of subjects, mean, and standard deviation, minimum, median and maximum) for continuous endpoints, and frequency and percentage for categorical endpoints.

All statistical analyses will be conducted using SAS<sup>®</sup>, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM, Version 3.2) implementation for human clinical trials and ADaM (Analysis Dataset Model, Version 1.0).

The treatments for all outputs will be labeled as and presented in the order below:

| GSP 301 placebo NS pH |
|-----------------------|
| GSP 301 placebo NS pH |
| GSP 301 NS |

The following conventions are applied to all data presentations and summaries:

#### Descriptive statistics

Minimum, Maximum: the same number of decimal places as the raw data Arithmetic mean, Standard Deviation (SD), Median: 1 more decimal place than the raw data.

Descriptive statistics will be presented aligned by decimal point.

#### Categorical Variables

The number and percentage of the responses are presented in the form xxx (xx.x)

Percentages: 1 decimal place

No display of percentage in case that number of subject is zero unless otherwise stated

#### P-values

3 decimal places

If the p-value is less than 0.001 then it will be presented as <0.001. If the rounded result is a value of 1.000, it will be displayed as >0.999




• Confidence Interval (CI) limits

The same decimal places as the estimate (in the case of mean, 1 more decimal place than the raw data, and in the case of percentage, 1 decimal place)

A table, figure, listing is to be generated for any required item where no data is available or reported. This will ensure to the health authorities that the tables, figures, listings and narratives are accounted for.

- Generate a table or listing which states "No Data Available" or "No Data Reported"
- Print a one line message indicating there was no report data available: "NO DATA AVAILABLE FOR THIS REPORT"

#### 12.1 Study Population Analyses

#### 12.1.1 Overview of Planned Analyses

The study population analyses will be based on the safety analysis set, unless otherwise specified. **Table 1** provides an overview of the planned study population analyses.




04-Apr-2017

**Table 1: Overview of Planned Study Population Analyses** 

| Display Type Data Displays Gene | | nerated | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject disposition | | | |
| Total screened | Y[1] | | |
| Treated with study medication during run-in period | Y[1] | | |
| Randomized | Y[2] | | |
| Study completion/withdrawal | Y[2] | | Υ |
| Reason for early termination | Y[2] | | Υ |
| Protocol Deviations | | | |
| Protocol deviations recorded in the eCRF | Y[2] | | Υ |
| Subjects included in /excluded from analysis population | tions | | |
| Summary of subjects in analysis population | Y[2] | | |
| Subjects excluded from each analysis populations | | | Υ |
| Subjects who withdrew due to inclusion/exclusion | | | Υ |
| criteria with number | | | ī |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | Y[3] | | Υ |
| Medical History | | | Υ |
| Exposure and Treatment Compliance | | | |
| Exposure | Y[2] | | Υ |
| Treatment Compliance | Y[2] | · | Υ |
| Concomitant Medications | | | |
| Prior Medications | | | Υ |
| Concomitant Medications | | | Υ |

#### NOTES:

- Y = Yes display generated.
- [1]: Data from clinic or database
- [2]: Display will be based on the SAS
- [3]: Display will be based on the SAS population and repeated for the FAS, PPS

#### 12.1.2 Supplementary Information for Study Population Tables and Listings

#### 12.1.2.1 Subject Disposition

The subject accountability and disposition information will be summarized by study treatment group. The number of subjects screened, treated with study medication during the run-in period, randomized, treated with study medication following randomization, and the number of subjects in each analysis set will be tabulated. In addition, completion status and primary reason for withdrawal will be summarized by study treatment group.




#### 12.1.2.2 Demographic and Other Baseline Characteristics

Demographics and other baseline characteristics will be summarized by treatment group separately for the SAS, FAS, PPS, and RQLQ(S) analysis set.

Continuous variables such as age will be summarized using descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum). Categorical variables such as sex and race will be summarized using frequencies and percentage.

All data will be listed by treatment and subject.

#### 12.1.2.3 Medical History

All relevant medical and surgical history and current medical conditions will be recorded at the Screening Visit (Visit 1).

Medical history data will be listed by treatment and subject.

#### 12.1.2.4 Extent of Exposure

The number of subjects exposed to each study treatment will be summarized.

The number of days on treatment and the number of days on study will be summarized by study treatment.

Treatment compliance will be calculated as follows:

Compliance = (the total number of doses actually taken) / (total number of doses scheduled)\*100 where:

For subjects who have completed the study, the total number of doses scheduled is 728 (2\*7\*52=728, for 52 weeks).

For subjects whose participation is terminated early, compliance will be determined from their duration in the study, up to the time they are considered early terminated. The total number of doses scheduled = the minimum between 728 and [(Date of Discontinuation – Date of First Application +1)\*2].

Subjects taking fewer than 75% or more than 125% of the required doses will be considered non-compliant with dosing.

In addition, treatment compliance will be classified into four categories (less than 75%, 75% to 100%, greater than 100% to125%, and greater than 125%). Treatment compliance will be summarized by categories and study treatment.

#### 12.1.2.5 Concomitant Medications

At Visit 1 subjects will be questioned about current and prior concomitant medication use. At other visits subjects will be questioned about ongoing or new concomitant medication use.

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|




Medications will be grouped and presented as follows:

- Prior medications: defined as medications that started and ended before the first administration of the study medication.
- Concomitant medications: defined as medications either ongoing or ended on or after the first dose of study medication.

All prior and concomitant medications taken since screening until the end of the study will be listed by treatment and subject.

- If the end date and 'ongoing' are missing then the medication will be considered as concomitant medication.
- In cases of partial end dates, the following conventions will be applied:
  - If the end day is missing, and the end month and year are not missing, the end day will be imputed using the last day of the month.
  - If the end day and month is missing, and the end year is not missing, the end day and month will be imputed using '31DEC'. If this leads to a date after the last visit date, then the last visit date will be used instead.
  - If the end date is completely missing, the end date will be imputed using the last visit date.
- The partial dates will be provided as such in the subject data listings (with the imputed dates).

#### 12.2 Safety Analyses

#### 12.2.1 Overview of Planned Safety Analyses

The safety analyses will be based on the SAS, unless otherwise specified.

Table 2 provides an overview of the planned analyses.




04-Apr-2017

Table 2: Overview of Planned Safety Analyses

| Display Type | Data Displays Generated | | rated |
|---------------------------------|-------------------------|--------|---------|
| | Table | Figure | Listing |
| Adverse Events | | | |
| Overview | Y[2] | | |
| Treatment Emergent AEs | Y[1][2] | | Υ |
| Treatment Emergent AEs Severity | Y[2] | | Υ |
| Drug-Related AEs | Y[2] | | Υ |
| Placebo Run-In Period AEs | Y[2] | | Υ |
| AEs Leading to Withdrawal | | | Υ |
| SAEs | Y[2] | | Υ |
| Treatment Emergent SAEs | Y[2] | | Υ |
| Laboratory | | | |
| Biochemistry | Y[3] [2] | | Υ |
| Haematology | Y[3] [2] | | Υ |
| Urinalysis | Y[3] [2] | | Υ |
| Pregnancy Test Results | | | Υ |
| Other | | | |
| Vital Signs | Y[4] [2] | | Υ |
| ECGs | Y [5] [2] | | Υ |
| Physical Examination | Y[6] [2] | | Y |
| Focused ENT Examination | Y[7] [2] | | Υ |

#### NOTES:

- Y = Yes display generated.
- [1]: Display will also be produced by SOC, severity, and by relationship to study medication
- [2]: Display will be based on safety analysis set
- [3]: Display will be produced separately for overall laboratory assessments (inc. change from baseline), change from baseline in laboratory results, and potentially clinically significant laboratory results, and shift tables
- [4]: Display will be produced separately for overall summary (inc. change from baseline), for potentially clinically significant results, and shift tables
- [5]: Display will be produced separately for overall summary (inc. change from baseline), change from baseline in ECG interpretation, and potentially clinical significant ECGs, and shift tables
- [6]:Display will be produced separately for overall summary, and for potentially clinically significant results
- [7]:Display will be produced separately for overall summary, and for




| Display Type | Data Displays Generated | | |
|--------------|-------------------------|--------|---------|
| | Table | Figure | Listing |

potentially clinically significant results

#### 12.2.2 Adverse Events

All AEs will be coded according to the current version of MedDRA (version 18.1 or later). Adverse events occurring between the subjects signing informed consent and administration of the first dose of the randomized study medication will be regarded as pre-treatment AEs and will be included in the subject listings but not in the summary tables. Adverse events occurring after the first dose of the randomized study medication will be defined as treatment-emergent adverse events (TEAEs) and will be listed and summarized by System Organ Class (SOC) and Preferred Term (PT).

The safety endpoints related to AEs are:

- Proportion of subjects with TEAEs.
- Proportion of subjects with treatment-related TEAEs.
- Incidence, type, and severity of the TEAEs after 30 weeks of study treatment.
- Incidence, type, and severity of the TEAEs after 52 weeks of study treatment.

Summaries of the number and percentage of subjects with TEAEs and the number of TEAEs experienced will be presented by treatment group. The number of subjects and the number of TEAEs will be presented using frequency counts and percentages, overall and by SOC and PT. The percentages will be calculated as the number of subjects with TEAEs divided by the number of subjects in the safety analysis set. Tables of the number and percentage of subjects and the number of TEAEs by intensity and by relationship to study medication will also be presented. Similar tables will be created for treatment related AEs. Events will be assigned to the study treatment administered prior to the start of the TEAE. Events that occurred during discharge and final follow-up will be assigned to the final treatment.

The number and percentage of subjects with a TEAE that has a start date within 30 weeks of the start of treatment (≤182 days) will be summarized by severity and study treatment group, overall, and by SOC and PT using frequency counts and percentages. A similar summary will be produced including all TEAEs during the study (i.e., after 52 weeks of treatment).

The overall p-value of the comparison among three treatment groups by SOC and PT will be produced using Fisher's exact test for each SOC and PT as well as overall subjects with at least one TEAEs.




04-Apr-2017

Additionally, the number and percentage of AEs, SAEs, TEAEs leading to discontinuation, and TEAEs related to the IP will be summarized by SOC, PT, and study treatment group.

#### 12.2.3 Adverse Events of Special Interest (AESI)

The following SOC terms will be grouped into a Special Interest AE Group.

| Special<br>Interest AE<br>Group | SOCs | PTs |
|---|---|---|
| | Respiratory, thoracic and mediastinal disorders | Nasal septum perforation |
| Nasal<br>toxicities | Respiratory, thoracic and mediastinal disorders | Nasal mucosal ulcer |
| | Respiratory, thoracic and mediastinal disorders(Primary) | Epistaxis |
| On the almaid | Eye disorders | -Open angle glaucoma<br>-Glaucoma |
| Opthalmic toxicities | Investigations | Intraocular pressure increased |
| | Eye disorders | Cataract |
| Somnolence | Nervous system disorders(Primary) | Somnolence |
| Others | Nervous system disorders (Primary) | Dysgeusia |
| Olliers | Nervous system disorders | Headaches |

The following tables will be produced for AESI:

- Summary of Treatment Emergent Adverse Events of Special Interest (Safety Analysis Set)
- Summary of Treatment Related Emergent Adverse Events of Special Interest (Safety Analysis Set)
- Summary of Treatment Emergent Adverse Events of Special Interest by Severity (Safety Analysis Set)
- Summary of Treatment Emergent Adverse Events of Special Interest by Relationship to Study Treatment (Safety Analysis Set)

## 12.2.4 Laboratory Data

Clinical laboratory test data (hematology, biochemistry, and urinalysis), will be summarized for each visit at which laboratory assessments are done (Screening Visit [Visit 1], Week 30 [Visit 8], and Week 52 [Visit 12]).




Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) will be presented for laboratory data as well as change from baseline by treatment and visit.

Baseline is defined as the last available lab values at Screening Visit [Visit 1].

In addition, values outside the normal range and values deemed as clinically significant by the Investigator will be listed. The number of subjects with values of potentially clinical significance determined by the investigator will be tabulated by treatment group and visit.

Shift tables will present changes from baseline in laboratory data (categorized as normal; abnormal, not clinically significant; and abnormal, clinically significant) to end of treatment.

All laboratory data will be listed by treatment and subject.

#### 12.2.5 Pregnancy Test

All females of child bearing potential will have a urine pregnancy test at each visit.

Pregnancy test results will be listed by treatment and subject.

#### 12.2.6 Vital Signs

Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) will be used to summarize vital sign results and changes from baseline by treatment group and time point (Week 1 [Visit 2], Week 30 [Visit 8] and Week 52 [Visit 12]).

Baseline is defined as the last available vital signs at Randomization Visit [Visit 2].

Values outside the respective normal range and values deemed as clinically significant by the Investigator will be listed.

The number of subjects with values of potential clinical significance determined by the investigator will be tabulated by treatment group and visit.

Shift tables will present changes from baseline in vital signs (categorized as normal; abnormal, not clinically significant; and abnormal, clinically significant) to end of treatment.

All vital sign data will be listed by treatment and subject.

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|




#### 12.2.7 ECGs

Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) for ECG parameters and changes from baseline will be presented by treatment group.

Baseline is defined as the last available ECG values at Screening Visit [Visit 1].

Shift tables will present changes from baseline in ECG interpretation (categorized as normal; abnormal, not clinically significant; and abnormal, clinically significant) to end of treatment.

The number of subjects with values of potential clinical significance determined by the investigator will be tabulated by treatment group and visit.

All ECG data will be listed by treatment and subject.

#### 12.2.8 Physical Examinations

Descriptive statistics (frequency and percentage) will be used to summarize physical examination results by treatment group and time point (Screening Visit, Week 30 and Week 52).

In addition, the number of subjects with values of potential clinical significance determined by the investigator will be tabulated.

All physical examination data will be listed by treatment and subject.

#### 12.2.9 ENT examination

Descriptive statistics (frequency and percentage) will be used to summarize ENT examination results by treatment group and time point (Screening Visit, Week 30 and Week 52).

In addition, the number of subjects with values of potential clinical significance determined by the investigator will be tabulated.

All ENT examination data will be listed by treatment and subject.

#### 12.2.10 Rescue Medication



Protocol Number: GPL/CT/2014/018/III SAP Version Number: Version 1.0


(Study No. GSP 301-303)

Descriptive statistics will be used to summarize the number and percentage of subjects who used rescue medication by treatment and rescue medication categories.

Rescue medication along with the type, dose, and duration of rescue medication will be listed by treatment and subject.

#### 12.3 Efficacy Analyses of Efficacy Endpoints

For all efficacy statistical analysis of efficacy endpoints, the comparison of interest will be GSP 301 NS vs. placebo NS pH The statistical analysis will only include up to week 52 data in the analysis.

#### 12.3.1 Overview of Efficacy Analysis of the Efficacy Endpoints (rTNSS, iTNSS, RQLQ(S) over the first 6, 30, and 52 weeks of treatment)

The efficacy analysis of the efficacy endpoints will be performed on the FAS (primary) and the PPS (supportive) for rTNSS and iTNSS. For RQLQ(S) outputs will be performed on the FAS.

Table 3 provides an overview of the planned efficacy analyses.




04-Apr-2017

#### **Table 3: Overview of Planned Efficacy Analyses**

| | Sta | | Sun | nmary | Individual |
|---|---|---|---|---|---|
| | Analy | 1 | | | |
| | Т | F | Т | F | L |
| Change from baseline in the average AM rTNSS ov treatment | er the firs | st 6, 30 | , and t | 52 wee | ks of |
| rTNSS – MMRM – FAS | Υ | Υ | | | |
| rTNSS – MMRM – PPS | Υ | Υ | | | |
| rTNSS Raw Data | | | | | |
| By Day (including post-baseline and change from | | | | | Y |
| baseline) - SAS | | | | | |
| Change from baseline in the average AM iTNSS over the first 6, 30, and 52 weeks of | | | | | |
| treatment | | | | | |
| iTNSS - MMRM - FAS | Υ | Υ | | | |
| iTNSS - MMRM - PPS | Υ | Υ | | | |
| iTNSS Raw Data | | | | | |
| By Day (including post-baseline and change from | | | | | Y |
| baseline) - SAS | | | | | |
| Change from baseline in the overall RQLQ(S) score | at Week | s 6, 30 | , and | 52 | |
| RQLQ(S) – MMRM – FAS | Υ | Υ | Υ | | |
| RQLQ(S) Raw Data | | | | | |
| Visit (including post-baseline and change from | | | | | Υ |
| baseline) - SAS | | | | | |
| NOTES: | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TF related to any formal statistical analyses (i.e. modeling) conducted.
- Summary = Represents TF related to summaries (i.e. descriptive statistics) of the baseline, post-treatment and change from baseline for the primary efficacy analyses method.
- Individual = Represents L related to any displays of individual subject observed raw data.

# 12.3.2 Analysis Method of the Efficacy Endpoints (rTNSS, iTNSS, RQLQ(S)): Mixed Model Repeated Measures Approach

# 12.3.2.1 Change from baseline in the average AM rTNSS over the first 6, 30 and 52 weeks of treatment

The efficacy endpoints rTNSS will be analyzed using a mixed model repeated measures model, adjusting for covariates that include treatment, site, baseline and week as the within-subject effect (for both the FAS and the PPS). The interactions of

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|




04-Apr-2017

site-by-treatment and baseline-by-treatment will be investigated separately in the model and will only be included in final model if they are statistically significant at the alpha=5% level. An unstructured (UN) covariance will be assumed. If the model does not converge using the unstructured covariance structure, the autoregressive (order 1) AR(1) structure will be used. If this also does not converge other covariance structures deemed appropriate to fit the data will be used. This method will assume that any missing data is Missing at Random (MAR). The statements of a SAS PROC MIXED analysis would be (if the interactions of treatment\*baseline and treatment\*site is not statistically significant):

proc mixed; class subject treatment site week: model change = treatment site baseline week; repeated week / subject = subject type=UN; Ismeans treatment / cl diff e; ods output Ismeans=Ismeans: ods output diffs=diffs; run ; quit ;

The adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with 95% confidence intervals for the differences and p-values for the treatment comparisons. The adjusted means and estimated treatment differences for the treatment comparisons will also be plotted, with corresponding 95% confidence intervals.

The responses for the first 6, 30 and 52 weeks of treatment will all be analysed in separate statistical models.

A multiple, imputation-based approach may be considered for handling missing data for AM rTNSS upon review of amount of missing data observed.

#### 12.3.2.2 Change from baseline in the average AM iTNSS over the first 6, 30 and **52** weeks of treatment

AM iTNSS will be analyzed using same methods as described in Section 12.3.2.1.

The efficacy endpoints iTNSS will be analyzed using a mixed model repeated measures model, adjusting for covariates that include treatment, site, baseline and week as the within-subject effect (for both the FAS and the PPS). The interactions of site-by-treatment and baseline-by-treatment will be investigated separately in the model and will only be included in final model if they are statistically significant at the alpha=5% level. An unstructured (UN) covariance will be assumed. If the model does not converge using the unstructured covariance structure, the autoregressive (order 1) AR(1) structure will be used. If this also does not converge other covariance structures deemed appropriate to fit the data will be used. This method will assume that any missing data is Missing at Random (MAR). The statements of a



Protocol Number: GPL/CT/2014/018/III (Study No. GSP 301-303)

run; quit;

SAP Version Number:


SAS PROC MIXED analysis would be (if the interactions of treatment\*baseline and treatment\*site is not statistically significant):

proc mixed; class subject treatment site week; model change = treatment site baseline week; repeated week / subject = subject type=UN; Ismeans treatment / cl diff e; ods output Ismeans=Ismeans; ods output diffs=diffs;


The adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with 95% confidence intervals for the differences and p-values for the treatment comparisons. The adjusted means and estimated treatment differences for the treatment comparisons will also be plotted, with corresponding 95% confidence intervals.

The responses for the first 6, 30 and 52 weeks of treatment will all be analysed in separate statistical models.

A multiple, imputation-based approach may be considered for handling missing data for AM iTNSS upon review of amount of missing data observed.

#### 12.3.2.3 Change from baseline in the overall RQLQ(S) score at Weeks 6, 30, and 52

RQLQ(S) (for the FAS) will be analyzed using similar methods as described in Section 12.3.2.1, with the following differences:

- Interaction of week-by-treatment will be included in the statistical model
  - Addition of week\*treatment interaction in SAS model statement
  - Week\*treatment interaction stated in SAS Ismeans statement.
- The responses at 6, 30 and 52 weeks of treatment will all be analysed in the same statistical model.

The interactions of site-by-treatment and baseline-by-treatment will be investigated separately in the model and will only be included in final model if they are statistically significant at the alpha=5% level. An unstructured (UN) covariance will be assumed. If the model does not converge using the unstructured covariance structure, the autoregressive (order 1) AR(1) structure will be used. If this also does not converge other covariance structures deemed appropriate to fit the data will be used.

For each visit, the adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with 95% confidence intervals for the differences and p-values for the treatment comparisons.




The adjusted means and estimated treatment differences for the treatment comparisons will also be plotted, with corresponding 95% confidence intervals.

#### 12.3.6 Examination of Subgroups

As well as producing summary tables for the efficacy endpoints rTNSS and iTNSS, the following subgroups of clinical interest will also be summarized for the FAS only by treatment group and week: age group (12-17, 18-65, 65 and above), sex (female/male), race (American Indian or Alaska Native, Asian, Black/African American, Other and White) and ethnicity (Hispanic or Latino and Not Hispanic or Latino).

#### 12.4 Efficacy Analyses of Other Efficacy Endpoints

#### 12.4.1 Overview of Analysis of the Other Efficacy Endpoints

The efficacy analysis of the other efficacy endpoints will be performed on the FAS only, unless otherwise specified. For RQLQ(S) certain outputs will also be performed on the RQLQ(S) analysis set. The interaction of site-by-treatment and baseline-by-treatment will not be investigated for the other efficacy endpoints.

Efficacy analyses of other efficacy endpoints include the following:

#### **Nasal symptoms:**

- Change from baseline in the average AM subject-reported reflective individual nasal symptoms over the first 6, 30, and 52 weeks of treatment.
- Change from baseline in the average AM subject-reported instantaneous individual nasal symptoms over the first 6, 30, and 52 weeks of treatment.
- Change in the average AM subject-reported rTNSS and iTNSS from baseline to the end of each treatment week.
- Change in the average AM subject-reported reflective individual nasal symptoms from baseline to the end of each treatment week.
- Change in the average AM subject-reported instantaneous individual nasal symptoms from baseline to the end of each treatment week.

Physician assessed Nasal Symptom Score (PNSS), Rhinoconjunctivitis Quality of Life Questionnaire – Standardized Activities (RQLQ(S)), and Rhinitis Control Assessment Test (RCAT):

- Change from baseline in PNSS and physician assessed individual nasal symptoms at Weeks 6, 30, and 52.
- Change from baseline in individual domains of the RQLQ(S) at Weeks 6, 30, and 52 for the FAS.

|---------------------------------------|----------------|
|---------------------------------------|----------------|



Protocol Number: GPL/CT/2014/018/III SAP Version Number: Version 1.0


(Study No. GSP 301-303)

• Change from baseline in overall RQLQ(S) score and individual domains of the RQLQ(S) at Weeks 6, 30, and 52 for the RQLQ(S) Analysis Set.

- Change from baseline in the RCAT at Weeks 6, 30, and 52.
- Change from baseline in individual domains of the RCAT at Weeks 6, 30, and 52.

Table 4 provides an overview of the planned efficacy analyses.




Table 4: Overview of Planned Efficacy Analyses for Other Efficacy Endpoints

| Table 4. Overview of Flatilied Efficacy | Stats Analysis Summary Individual | | | | |
|---|---|---|---|---|---|
| | | | _ | mmary | Individual |
| | T | F | T | F | L |
| Change from baseline in the average AM reflective individual nasal symptoms | | | | | |
| over the first 6, 30, and 52 weeks of treatment | | | | | |
| MMRM – FAS | Υ | | | | Υ |
| Change from baseline in the average AM instantaneous individual nasal | | | | | |
| symptoms over the first 6, 30, and 52 weeks of treatment | | | | | |
| MMRM – FAS | Υ | | | | Υ |
| Change in the average AM subject-reported rTNSS and iTNSS from baseline to | | | | | |
| the end of each treatment week | | | | | |
| rTNSS – MMRM – FAS | Υ | | Υ | | Y |
| rTNSS - PPS | | | Υ | | |
| iTNSS – MMRM – FAS | Υ | | Υ | | Υ |
| iTNSS - PPS | | | Υ | | |
| Change in the average AM reflective individual nasal symptoms from baseline to | | | | | |
| the end of each treatment week | | | | | |
| MMRM – FAS | Y | | Υ | | Υ |
| Change in the average AM instantaneous individual nasal symptoms from | | | | | |
| baseline to the end of each treatment week | | | | | |
| MMRM – FAS | Υ | | Υ | | Υ |
| Change from baseline in PNSS and physician assessed individual nasal | | | | | |
| symptoms at Weeks 6, 30, and 52 | | | | | |
| MMRM – FAS | Υ | | Υ | | Υ |
| Change from baseline in individual domains of the RQLQ(S) at Weeks 6, 30, and | | | | | |
| 52 for the FAS | | | | | |
| MMRM – FAS | Υ | | Υ | | Y |
| Change from baseline in overall RQLQ(S) score and individual domains of the | | | | | |
| RQLQ(S) at Weeks 6, 30, and 52 for the RQLQ(S) Analysis Set | | | | | |
| MMRM – RQLQ analysis set | Y | | Υ | | |
| Change from baseline in the RCAT at Weeks 6, 30, and 52 | | | | | |
| MMRM – FAS | Υ | | Υ | | Υ |
| Change from baseline in individual domains of the RCAT at Weeks 6, 30, and 52 | | | | | |
| MMRM – FAS | Υ | | Υ | | Y |
| NOTES: | 1 | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TF related to any formal statistical analyses (i.e. modeling) conducted.
- Summary = Represents TF related to summaries (i.e. descriptive statistics) of the baseline, post-treatment and change from baseline for the primary efficacy analyses method.
- Individual = Represents L related to any displays of individual subject observed raw data.




#### 12.4.2 Analysis of Change from Baseline in Other Efficacy Endpoints

# 12.4.2.1 Change from baseline in the average AM reflective and AM instantaneous individual nasal symptoms over the first 6, 30, and 52 weeks of treatment

Similar to the analysis mentioned in section 12.3.2.1, the endpoints will be analyzed separately using a mixed model repeated measures model (by each individual nasal symptom), adjusting for covariates that include treatment, site, baseline and week as the within-subject effect (for the FAS). An unstructured (UN) covariance will be assumed. If the model does not converge using the unstructured covariance structure, the autoregressive (order 1) AR(1) structure will be used. If this also does not converge other covariance structures deemed appropriate to fit the data will be used. The statements of a SAS PROC MIXED analysis would be:

proc mixed;

by individual nasal symptom; class subject treatment site week; model change = treatment site baseline week; repeated week / subject = subject type=UN; Ismeans treatment / cl diff e; ods output Ismeans=Ismeans; ods output diffs=diffs; run; quit;

For each individual nasal symptom, the adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with 95% confidence intervals for the differences and p-values for the treatment comparisons. The adjusted means and estimated treatment differences for the treatment comparisons will also be plotted, with corresponding 95% confidence intervals.

The responses for the first 6, 30 and 52 weeks of treatment will all be analysed in separate statistical models.

# 12.4.2.2 Change in the average AM subject-reported rTNSS and iTNSS from baseline to the end of each treatment week

The efficacy endpoints rTNSS and iTNSS will be analyzed separately using a mixed model repeated measures model, adjusting for covariates that include treatment, site, baseline and week as the within-subject effect, and the model will include treatment\*week interaction term (for the FAS). The statements of a SAS PROC MIXED analysis would be:

proc mixed;




class subject treatment site week;
model change = treatment site baseline week treatment\*week;
repeated week / subject = subject type=UN;
Ismeans treatment treatment\*week / cl diff e;
ods output Ismeans=Ismeans;
ods output diffs=diffs;
run; quit;

For each week, the adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with 95% confidence intervals for the differences and p-values for the treatment comparisons. The adjusted means and estimated treatment differences for the treatment comparisons will also be plotted, with corresponding 95% confidence intervals.

Descriptive statistics (number of subjects, mean, standard deviation, median, minimum and maximum) will be provided for baseline, post treatment and change from baseline by treatment group and week (for both the FAS and the PPS).

# 12.4.2.3 Change in the average AM reflective and AM instantaneous individual nasal symptoms from baseline to the end of each treatment week

Similar to Section 12.4.2.2, the efficacy endpoints will be analyzed separately using a mixed model repeated measures model, adjusting for covariates that include treatment, site, baseline and week as the within-subject effect, and the model will include treatment\*week interaction term (for the FAS). The statements of a SAS PROC MIXED analysis would be:

proc mixed;

by individual nasal symptom; class subject treatment site week; model change = treatment site baseline week treatment\*week; repeated week / subject = subject type=UN; Ismeans treatment treatment\*week / cl diff e; ods output lsmeans=Ismeans; ods output diffs=diffs; run; quit;

For each individual symptom and each week, the adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with 95% confidence intervals for the differences and p-values for the treatment comparisons. The adjusted means and estimated treatment differences for the treatment comparisons will also be plotted, with corresponding 95% confidence intervals.




12.4.2.4 Change from baseline in PNSS, Overall RQLQ(S) score and RCAT at Weeks 6, 30, and 52

RQLQ(S) (for RQLQ(S) Analysis Set), PNSS (for FAS) and RCAT (for FAS) will be analyzed separately using the same methods as described in Section 12.3.2.2 with the exeption that the interaction of site-by-treatment and baseline-by-treatment will not be investigated separately in the model.

12.4.2.5 Change from baseline in physician assessed individual nasal symptoms, individual domains of the RQLQ(S) and individual domains of the RCAT at Weeks 6, 30, and 52

RQLQ(S) (for both the FAS and RQLQ(S) Analysis Set), PNSS (for FAS) and RCAT (for FAS) will be analyzed separately using the same methods as described in Section 12.4.2.4, with the addition of a by statement (for the individual symptoms/domains) in the SAS PROC MIXED model.




#### Appendix 1

The following shells are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. Additional Tables, Listings and Figures will be generated, as needed, following the data analysis (post-hoc). All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or later, unless otherwise noted. In general, Listings will be sorted and presented by treatment and subject number. Subject number when broken down consists of the Site Number and Subject Number.




04-Apr-2017

#### Tables:

- T14.1.9.1 Summary of Subject Disposition
- T14.1.9.2.1 Summary of Protocol Deviations During Randomized Treatment Period (Safety Analysis Set)
- T14.1.9.2.2 Summary of Protocol Deviations during Placebo Run-In Period
- T14.1.9.2.3 Summary of Major Protocol Deviations during Randomized Treatment Period
- T14.1.9.3 Summary of Subjects in Each Analysis Set
- T14.1.9.4.1 Summary of Demographic Data (Safety Analysis Set)
- T14.1.9.4.2 Summary of Demographic Data (Full Analysis Set)
- T14.1.9.4.3 Summary of Demographic Data (Per Protocol Set)
- T14.1.9.4.4 Summary of Demographic Data (RQLQ(S) Analysis Set)
- T14.1.9.5.1 Overall Summary of Treatment Emergent Adverse Events after 52 Weeks of Study

  Treatment (Safety Analysis Set)
- T14.1.9.5.2 Overall Summary of Treatment Emergent Adverse Events after 30 Weeks of Study Treatment (Safety Analysis Set)
- T14.1.9.5.3 Summary of Treatment Emergent Adverse Events after 52 Weeks of Study Treatment (Safety Analysis Set)
- T14.1.9.5.4 Summary of Treatment Emergent Adverse Events after 30 Weeks of Study Treatment (Safety Analysis Set)
- T14.1.9.5.5 Summary of Treatment-Related Emergent Adverse Events after 52 Weeks of Study Treatment (Safety Analysis Set)
- T14.1.9.5.6 Summary of Treatment-Related Emergent Adverse Events after 30 Weeks of Study

  Treatment (Safety Analysis Set)
- T14.1.9.5.7 Summary of Treatment Emergent Adverse Events of Special Interest (Safety Analysis Set)
- T14.1.9.5.8 Summary of Treatment Related Emergent Adverse Events of Special Interest (Safety Analysis Set)
- T14.1.9.5.9 Summary of Treatment Emergent Adverse Events after 52 Weeks of Study
  Treatment by Severity (Safety Analysis Set)
- T14.1.9.5.10 Summary of Treatment Emergent Adverse Events after 30 Weeks of Study
  Treatment by Severity (Safety Analysis Set)
- T14.1.9.5.11 Summary of Treatment Emergent Adverse Events of Special Interest by Severity (Safety Analysis Set)
- T14.1.9.5.12 Summary of Treatment Emergent Adverse Events after 52 Weeks of Study
  Treatment by Relationship to Study Treatment (Safety Analysis Set)
- T14.1.9.5.13 Summary of Treatment Emergent Adverse Events after 30 Weeks of Study
  Treatment by Relationship to Study Treatment (Safety Analysis Set)
- T14.1.9.5.14 Summary of Treatment Emergent Adverse Events of Special Interest by Relationship to Study Treatment (Safety Analysis Set)
- T14.1.9.5.15 Summary of Treatment Emergent Serious Adverse Events after 52 Weeks of Study Treatment (Safety Analysis Set)
- T14.1.9.5.16 Summary of Treatment Emergent Serious Adverse Events after 30 Weeks of Study Treatment (Safety Analysis Set)



T14.1.9.5.17 Summary of Treatment Related Emergent Serious Adverse Events after 52
Weeks of Study Treatment (Safety Analysis Set)

T14.1.9.5.18 Summary of Treatment Related Emergent Serious Adverse Events after 30
Weeks of Study Treatment (Safety Analysis Set)

T14.1.9.5.19.1 Overall Summary of Adverse Events During Placebo Run-In Period (Safety Analysis Set)

T14.1.9.5.19.2 Overall Summary of Adverse Events Pre-Randomization

T14.1.9.6.1 Summary of Clinical laboratory Assessment (Biochemistry) (Safety Analysis Set)

T14.1.9.6.2 Summary of Clinical laboratory Assessment (Hematology) (Safety Analysis Set)

T14.1.9.6.3 Summary of Clinical laboratory Assessment (Urinalysis) (Safety Analysis Set)

T14.1.9.6.4 Summary of Potentially Clinical Significant Laboratory Results (Biochemistry) (Safety Analysis Set)

T14.1.9.6.5 Summary of Potentially Clinical Significant Laboratory Results (Hematology) (Safety Analysis Set)

T14.1.9.6.6 Summary of Potentially Clinical Significant Laboratory Results (Urinalysis) (Safety Analysis Set)

T14.1.9.6.7 Shift Tables for Changes from Baseline in Laboratory Results (Biochemistry) to End of Treatment (Safety Analysis Set)

T14.1.9.6.8 Shift Tables for Changes from Baseline in Laboratory Results (Hematology) to End of Treatment (Safety Analysis Set)

T14.1.9.6.9 Shift Tables for Changes from Baseline in Laboratory Results (Urinalysis) to End of Treatment (Safety Analysis Set)

T14.1.9.7.1 Summary of Vital Signs (Safety Analysis Set)

T14.1.9.7.2 Summary of Potentially Clinical Significant Vital Signs (Safety Analysis Set)

T14.1.9.7.3 Shift Tables for Changes from Baseline in Vital Signs to End of Treatment (Safety Analysis Set)

T14.1.9.8.1 Summary of ECGs (Safety Analysis Set)

T14.1.9.8.2 Summary of Potentially Clinical Significant ECGs (Safety Analysis Set)

T14.1.9.8.3 Shift Tables for Changes from Baseline in ECG Interpretation to End of Treatment (Safety Analysis Set)

T14.1.9.9 Summary of Physical Examinations (Safety Analysis Set)

T14.1.9.10.1 Summary of Focused ENT Examination (Safety Analysis Set)

T14.1.9.10.2 Summary of Potentially Clinical Significant Focused ENT Examination (Safety Analysis Set)

T14.1.9.11.1 Summary of Extent of Exposure during the Post Randomization Treatment Period (Safety Analysis Set)

T14.1.9.11.2 Summary of Rescue Medication (Safety Analysis Set)

T14.1.9.12.1 Summary of Average AM rTNSS (Full Analysis Set)

T14.1.9.12.2 Summary of Repeated Measures Analysis Results in Average AM rTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)

T14.1.9.12.3 Summary of Average AM rTNSS (Per Protocol Set)

T14.1.9.12.4 Summary of Repeated Measures Analysis Results in Average AM rTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set)




04-Apr-2017

- T14.1.9.12.5 Subgroup Analyses (Age Group): Summary of Average AM rTNSS (Full Analysis Set)
- T14.1.9.12.6 Subgroup Analyses (Sex): Summary of Average AM rTNSS (Full Analysis Set)
- T14.1.9.12.7 Subgroup Analyses (Race): Summary of Average AM rTNSS (Full Analysis Set)
- T14.1.9.12.8 Subgroup Analyses (Ethnicity): Summary of Average AM rTNSS (Full Analysis Set)
- T14.1.9.13.1 Summary of Average AM iTNSS (Full Analysis Set)
- T14.1.9.13.2 Summary of Repeated Measures Analysis Results in Average AM iTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)
- T14.1.9.13.3 Summary of Average AM iTNSS (Per Protocol Set)
- T14.1.9.13.4 Summary of Repeated Measures Analysis Results in Average AM iTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set)
- T14.1.9.13.5 Subgroup Analyses (Age Group): Summary of Average AM iTNSS (Full Analysis Set)
- T14.1.9.13.6 Subgroup Analyses (Sex): Summary of Average AM iTNSS (Full Analysis Set)
- T14.1.9.13.7 Subgroup Analyses (Race): Summary of Average AM iTNSS (Full Analysis Set)
- T14.1.9.13.8 Subgroup Analyses (Ethnicity): Summary of Average AM iTNSS (Full Analysis Set)
- T14.1.9.14.1 Summary of the Overall RQLQ(S) (Full Analysis Set)
- T14.1.9.14.2 Summary of Repeated Measures Analysis Results in Overall RQLQ(S) at Weeks 6, 30, and 52 (Full Analysis Set)
- T14.1.9.14.3 Summary of Overall RQLQ(S) (RQLQ(S) Analysis Set)
- T14.1.9.14.4 Summary of Repeated Measures Analysis Results in Overall RQLQ(S) at Weeks 6, 30, and 52 (RQLQ(S) Analysis Set)
- T14.1.9.15.1 Summary of Average AM Reflective Individual Nasal Symptoms (Full Analysis Set)
- T14.1.9.15.2 Summary of Repeated Measures Analysis Results in Average AM Reflective
  Individual Nasal Symptoms over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)
- T14.1.9.16.1 Summary of Average AM Instantaneous Individual Nasal Symptoms (Full Analysis Set)
- T14.1.9.16.2 Summary of Repeated Measures Analysis Results in Average AM Instantaneous
  Individual Nasal Symptoms over the First 6, 30, and 52 Weeks of Treatment (Full
  Analysis Set)
- T14.1.9.17.1 Summary of Repeated Measures Analysis Results in Average AM rTNSS over Each Treatment Week (Full Analysis Set)
- T14.1.9.17.2 Summary of Repeated Measures Analysis Results in Average AM iTNSS over Each Treatment Week (Full Analysis Set)
- T14.1.9.18.1 Summary of Repeated Measures Analysis Results in Average AM Subjectreported Reflective Individual Nasal Symptoms over Each Treatment Week (Full Analysis Set)
- T14.1.9.18.2 Summary of Repeated Measures Analysis Results in Average AM Subjectreported Instantaneous Individual Nasal Symptoms over Each Treatment Week (Full Analysis Set)
- T14.1.9.19.1 Summary of the Physician Assessed Nasal Symptom Score (PNSS) (Full Analysis Set)




T14.1.9.19.2 Summary of Repeated Measures Analysis Results in Physician Assessed Nasal Symptom Score (PNSS) at Weeks 6, 30, and 52 (Full Analysis Set)

T14.1.9.20.1 Summary of the Physician Assessed Individual Nasal Symptom Score (Full Analysis Set)

T14.1.9.20.2 Summary of Repeated Measures Analysis Results in Physician Assessed Individual Nasal Symptom Score at Weeks 6, 30, and 52 (Full Analysis Set)

T14.1.9.21.1 Summary of the Individual Domains of the RQLQ(S) (Full Analysis Set)

T14.1.9.21.2 Summary of Repeated Measures Analysis Results in the Individual Domains of the RQLQ(S) at Weeks 6, 30, and 52 (Full Analysis Set)

T14.1.9.21.3 Summary of the Individual Domains of the RQLQ(S) (RQLQ(S) Analysis Set)

T14.1.9.21.4 Summary of Repeated Measures Analysis Results in the Individual Domains of the RQLQ(S) at Weeks 6, 30, and 52 (RQLQ(S) Analysis Set)

T14.1.9.22.1 Summary of RCAT (Full Analysis Set)

T14.1.9.22.2 Summary of Repeated Measures Analysis Results in RCAT at Weeks 6, 30, and 52 (Full Analysis Set)

T14.1.9.23.1 Summary of the Individual Domains of the RCAT (Full Analysis Set)

T14.1.9.23.2 Summary of Repeated Measures Analysis Results in the Individual Domains of the RCAT at Weeks 6, 30, and 52 (Full Analysis Set)

#### Listings:

- L16.2.1 Listing of Subject Disposition (Safety Analysis Set)
- L16.2.2 Listing of Protocol Deviations (Safety Analysis Set)
- L16.2.3.1 Listing of Subjects Excluded from the Per Protocol Set
- L16.2.3.2 Listing of Subjects Excluded from the Full Analysis Set
- L16.2.3.3 Listing of Subjects Who Withdrew Due to Inclusion/Exclusion Criteria (Safety Analysis Set)
- L16.2.4.1 Listing of Demographic Data (Safety Analysis Set)
- L16.2.4.2 Listing of Medical History (Safety Analysis Set)
- L16.2.4.3 Listing of Concomitant Medication (Safety Analysis Set)
- L16.2.4.4 Listing of Rescue Medication (Safety Analysis Set)
- L16.2.4.5 Listing of Skin Prick Test and Allergy Testing (Safety Analysis Set)
- L16.2.5.1 Listing of Visit Date Information (Safety Analysis Set)
- L16.2.5.2 Listing of Study Compliance (Safety Analysis Set)
- L16.2.5.3 Listing of Extent of Exposure (Safety Analysis Set)
- L16.2.6.1 Listing of AM Reflective Nasal Symptom Scores (Safety Analysis Set)
- L16.2.6.2 Listing of AM Instantaneous Nasal Symptom Scores (Safety Analysis Set)
- L16.2.6.3 Listing of the Average AM Reflective Nasal Symptom Scores (Safety Analysis Set)
- L16.2.6.4 Listing of the Average AM Instantaneous Nasal Symptom Score (Safety Analysis Set)
- <u>L16.2.6.5 Listing of Change from Baseline of the Average AM Reflective Nasal Symptom</u> <u>Scores (Safety Analysis Set)</u>
- L16.2.6.6 Listing of Change from Baseline of the Average AM Instantaneous Nasal Symptom Scores (Safety Analysis Set)
- L16.2.6.7 Listing of Rhinoconjunctivitis Quality of Life (RQLQ(S)) (Safety Analysis Set)




- <u>L16.2.6.8 Listing of Rhinoconjunctivitis Quality of Life (RQLQ(S)) by Domain (Safety Analysis Set)</u>
- L16.2.6.9 Listing of Change from Baseline in Rhinoconjunctivitis Quality of Life (RQLQ(S)) by Domain (Safety Analysis Set)
- <u>L16.2.6.10 Listing of Physician Assessed Nasal Symptom Scores (PNSS) (Safety Analysis Set)</u>
- L16.2.6.11 Listing of Change from Baseline in Physician Assessed Nasal Symptom Scores (PNSS) (Safety Analysis Set)
- L16.2.6.12 Listing of Rhinitis Control Assessment Test (RCAT) (Safety Analysis Set)
- L16.2.6.13 Listing of Change from Baseline in Rhinitis Control Assessment Test (RCAT) (Safety Analysis Set)
- <u>L16.2.7.1 Listing of Treatment Emergent Adverse Events by Treatment During Randomized</u>
  <u>Treatment Period (Safety Analysis Set)</u>
- L16.2.7.2 Listing of Adverse Events During Placebo Run-in Period
- L16.2.7.3 Listing of Pre-Treatment Adverse Events (Safety Analysis Set)
- L16.2.8.1 Listing of Clinical Laboratory Test Results (Biochemistry) (Safety Analysis Set)
- L16.2.8.2 Listing of Clinical Laboratory Test Results (Hematology) (Safety Analysis Set)
- L16.2.8.3 Listing of Clinical Laboratory Test Results (Urinalysis) (Safety Analysis Set)
- L16.2.8.4 Listing of Pregnancy Test Results (Safety Analysis Set)
- L16.2.8.5 Listing of Vital Signs (Safety Analysis Set)
- L16.2.8.6 Listing of 12-Lead ECGs (Safety Analysis Set)
- L16.2.8.7 Listing of Physical Examination (Safety Analysis Set)
- L16.2.8.8 Listing of Focused ENT Examination (Safety Analysis Set)
- L16.2.8.9 Listing of Eye Examination (Safety Analysis Set)

#### Figures:

- F15.1.1 LS Means with 95% CIs of AM Average rTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)
- F15.1.2 LS Means with 95% Cls of AM Average rTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set)
- F15.1.3 LS Means with 95% CIs of AM Average iTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)
- F15.1.4 LS Means with 95% CIs of AM Average iTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set)
- F15.1.5 LS Means with 95% CIs of Overall RQLQ(S) at Weeks 6, 30, and 52 (Full Analysis Set)
- F15.2.1 Treatment Differences of LS Means with 95% CIs of AM Average rTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)
- F15.2.2 Treatment Differences of LS Means with 95% CIs of AM Average rTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set)
- F15.2.3 Treatment Differences of LS Means with 95% CIs of AM Average iTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)
- F15.2.4 Treatment Differences of LS Means with 95% CIs of AM Average iTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set)




3)

- <u>F15.2.5 Treatment Differences of LS Means with 95% CIs of Overall RQLQ(S) at Weeks 6, 30,</u> and 52 (Full Analysis Set)
- F15.3.1 LS Means with 95% CIs of Average AM rTNSS over each Treatment Week (Full Analysis Set)
- F15.3.2 LS Means with 95% CIs of Average AM iTNSS over each Treatment Week (Full Analysis Set)
- F15.4.1 Treatment Differences of LS Means with 95% Cls of AM Average rTNSS over each Treatment Week (Full Analysis Set)
- F15.4.2 Treatment Differences of LS Means with 95% Cls of AM Average iTNSS over each Treatment Week (Full Analysis Set)

Protocol Number: GPL/CT/2014/018/III (Study No. GSP 301-303)

SAP Version Number: Version 1.0


### T14.1.9.1 Summary of Subject Disposition

| Subjects | GSP 301 placebo | GSP 301 placebo | GSP 301 | |
|---|---|---|---|---|
| · | NS pĤ | NS pH | NS | Total |
| | (N=xxx) | (N=xxx) | (N=xxx) | (N=xxx) |
| | n (%) | n (%) | n (%) | n (%) |
| Total Screened | | | | XXX |
| Screen failures | | | | XXX |
| Treated in run-in period | | | | XXX |
| Randomized | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Randomized failures | | | | XXX |
| Terminated early | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Completed study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Early Termination Reason | | | | |
| Adverse Event | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Death | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Lack of efficacy | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Lost to follow-up | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Non-compliance with study drug | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Physician Decision | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Protocol Deviation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Pregnancy | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Study terminated by sponsor | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Withdrawal by subject | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Withdrawal by parent/guardian | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Withdrawal of consent | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Others | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Data source: xx

Created on: ddmmmyy hh:mm


| AD-BST-05.02 23-Jan-2015 |
|------------------------------------------------------|
|------------------------------------------------------|

| GPL/CT/2014/018/III | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
| (Study No. GSP 301-303) | | 1 |

# T14.1.9.2.1 Summary of Protocol Deviations During Randomized Treatment Period (Safety Analysis Set)

| | GSP 301 placebo<br>NS pH<br>(N=xxx) | GSP 301 placebo<br>NS pH<br>(N=xxx) | GSP 301<br>NS<br>(N=xxx) |
|---|---|---|---|
| | n (%) | n (%) | n (%) |
| Total Subjects with Protocol Deviations | xxx (xx.x) | xxx(xx.x) | xxx (xx.x) |
| Total Deviations | XXX | XXX | XXX |
| Restricted medication/procedure used for the treatment of seasonal allergic rhinitis | XXX | XXX | xxx |
| Restricted medication/procedure used for reasons other than the treatment of seasonal allergic rhinitis | XXX | XXX | XXX |
| Lost to follow up | XXX | XXX | XXX |
| Enrolled in error | XXX | XXX | XXX |
| Randomized in error | XXX | XXX | XXX |
| Non-compliance with study drug | XXX | XXX | XXX |
| Non-compliance with study procedure | XXX | XXX | XXX |
| Outside visit window | XXX | XXX | XXX |
| Visit procedure not completed per protocol | XXX | XXX | XXX |
| Dosing procedure non-compliance | XXX | XXX | XXX |
| Lost to follow up | XXX | XXX | XXX |
| TNSS ratings non-compliance | XXX | XXX | XXX |
| Other | XXX | XXX | XXX |

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number: | SAP Version Number: | SAP Version Date: |
|-------------------------|---------------------|-------------------|
| GPL/CT/2014/018/III | Version 1.0 | 04-Apr-2017 |
| (Study No. GSP 301-303) | , elsion 1.0 | 04-Apr-2017 |

**T14.1.9.2.2 Summary of Protocol Deviations during Placebo Run-In Period**Repeat of T14.1.9.2.1 for placebo Run-in period

**T14.1.9.2.3 Summary of Major Protocol Deviations during Randomized Treatment Period**Repeat of T14.1.9.2.1 for major protocol deviations in treatment period

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|
| GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | Version 1.0 | 04-Apr-2017 |

### T14.1.9.3 Summary of Subjects in Each Analysis Set

| Number of Subjects | GSP 301 placebo<br>NS pH | GSP 301 placebo<br>NS pH | GSP 301<br>NS | Overall (N=xxx) |
|---|---|---|---|---|
| • | (N=xxx | (N=xxx | (N=xxx) | n (%) |
| | n (%) | n (%) | n (%) | |
| Randomized | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Safety analysis set | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Did not take any study medication | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Full analysis set | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Did not have at least one post-baseline primary AM rTNSS assessment | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Per protocol set | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Subjects with Major protocol violation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ROLO(S) Analysis Set | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Data source: xx

Created on: ddmmmyy hh:mm


| AD-BST-05.02 23-Jan-2015 Confidential Page | ge 45 of 152 |
|--------------------------------------------|--------------|
|--------------------------------------------|--------------|

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 017pi 2017 |

T14.1.9.4.1 Summary of Demographic Data (Safety Analysis Set)

| | | GSP 301 placebo<br>NS pH<br>(N=xxx) | GSP 301 placebo<br>NS pH<br>(N=xxx) | GSP 301<br>NS<br>(N=xxx) | Overall (N=xxx) |
|---|---|---|---|---|---|
| Age | n | XXX | XXX | XXX | XXX |
| | Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| Race n (%) | White | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Asian | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | American Indian or Alaska Native | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Black/African American | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Native Hawaiian or other Pacific | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Islander | | | | |
| | Other | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Ethnicity n (%) | Hispanic or Latino | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| , , | Not Hispanic or Latino | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Sex n (%) | Male | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ` / | Female | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

N= number of subjects in the treatment group; n= number of subjects with data available; % is based on N in the treatment group

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|
| (Study No. GSP 301-303) | r |

T14.1.9.4.2 Summary of Demographic Data (Full Analysis Set) Repeat of T14.1.9.4.1 for FAS

T14.1.9.4.3 Summary of Demographic Data (Per Protocol Set) Repeat of T14.1.9.4.1 for PPS

T14.1.9.4.4 Summary of Demographic Data (RQLQ(S) Analysis Set)

Repeat of T14.1.9.4.1 for RQLQ(S) analysis set

| | SAP Version Number: | SAP Version Date: |
|-------------------------|---------------------|-------------------|
| (Study No. GSP 301-303) | | 04-11p1-2017 |

T14.1.9.5.1 Overall Summary of Treatment Emergent Adverse Events after 52 Weeks of Study Treatment (Safety Analysis Set)

| | GSP 301 placebo | GSP 301 placebo | GSP 301 |
|---|---|---|---|
| | NS pH | NS pĤ | NS |
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Subjects in Safety Analysis Set (N1) | XXX | XXX | XXX |
| Subjects with at least one TEAE (n1(%)) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Discontinued study drug due to above AE (n1(%)) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| TEAEs reported (N2) | xxx | xxx | XXX |
| Mild (n2(%)) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Moderate (n2(%)) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Severe (n2(%)) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Not Related (n2(%)) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Related (n2(%)) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Death (n2(%)) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Serious AE (n2(%)) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

### T14.1.9.5.2 Overall Summary of Treatment Emergent Adverse Events after 30 Weeks of Study Treatment (Safety Analysis Set)

Repeat of T14.1.9.5.1 for after 30 weeks of study treatment

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### T14.1.9.5.3 Summary of Treatment Emergent Adverse Events after 52 Weeks of Study Treatment (Safety Analysis Set)

| | | NS | 801 placebo<br>S pH | NS 1 | 1 placebo<br>pH<br>=xxx | | SSP 301<br>NS<br>N=xxx) | |
|---|---|---|---|---|---|---|---|---|
| Body System | MedDRA<br>Term | Events | Subjects<br>n(%) | Events | Subjects<br>n(%) | Events | Subjects<br>n(%) | Fisher's<br>P-value |
| Subjects with at least one AEs | Total | XXX | xxx (xx.x) | XXX | xxx (xx.x) | XXX | xxx (xx.x) | X.XXXX |
| Ear and labyrinth disorders | Ear pain etc. | XXX | xxx (xx.x) | XXX | xxx (xx.x) | XXX | xxx (xx.x) | x.xxxx |

etc.

N = Total number of subjects in each treatment group in the safety set; n = number of subjects with adverse events in each MedDRA term; Percentages are based on total number of subjects in the safety set within each treatment group.

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|
| (Study No. GSP 301-303) | r |

### T14.1.9.5.4 Summary of Treatment Emergent Adverse Events after 30 Weeks of Study Treatment (Safety Analysis Set)

Repeat of T14.1.9.5.3 for after 30 weeks of study treatment

### T14.1.9.5.5 Summary of Treatment-Related Emergent Adverse Events after 52 Weeks of Study Treatment (Safety Analysis Set)

Repeat of T14.1.9.5.3 for related TEAEs after 52 weeks of study treatment

### T14.1.9.5.6 Summary of Treatment-Related Emergent Adverse Events after 30 Weeks of Study Treatment (Safety Analysis Set)

Repeat of T14.1.9.5.3 for related TEAEs after 30 weeks of study treatment

### T14.1.9.5.7 Summary of Treatment Emergent Adverse Events of Special Interest (Safety Analysis Set)

Repeat of T14.1.9.5.3 for AESI

### T14.1.9.5.8 Summary of Treatment Related Emergent Adverse Events of Special Interest (Safety Analysis Set)

Repeat of T14.1.9.5.3 for related TEAEs of AESI

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

# T14.1.9.5.9 Summary of Treatment Emergent Adverse Events after 52 Weeks of Study Treatment by Severity (Safety Analysis Set)

| | | G | SP 301 placebo NS pH # of Events (N=xx) | | GSP 301 placebo NS pH # of Events (N=xx) | | GSP 301<br>NS<br># of Events<br>(N=xx) | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Body System | MedDRA Term | Mild<br>n(%) | Moderate<br>n(%) | Severe<br>n(%) | Mild<br>n(%) | Moderate<br>n(%) | Severe<br>n(%) | Mild<br>n(%) | Moderate<br>n(%) | Severe<br>n(%) |
| Total AEs | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ear and labyrinth disorders | Ear pain | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Total number of subjects in each treatment group in the safety set; n = number of subjects with adverse events in each MedDRA term; Percentages are based on total number of subjects in the safety set within each treatment group

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|-------------------------|---------------------|-------------------|
| GPL/CT/2014/018/III | Version 1.0 | |
| (Study No. GSP 301-303) | V C131011 1.0 | 04-Apr-2017 |

# T14.1.9.5.10 Summary of Treatment Emergent Adverse Events after 30 Weeks of Study Treatment by Severity (Safety Analysis Set)

Repeat of T14.1.9.5.9 for after 30 weeks of study treatment

T14.1.9.5.11 Summary of Treatment Emergent Adverse Events of Special Interest by Severity (Safety Analysis Set)

Repeat of T14.1.9.5.9 for AESI

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|
| (Study No. GSP 301-303) | 1 |

# T14.1.9.5.12 Summary of Treatment Emergent Adverse Events after 52 Weeks of Study Treatment by Relationship to Study Treatment (Safety Analysis Set)

| | | GSP 301 p | olacebo | GSP 301 | placebo | GSP | 301 |
|---|---|---|---|---|---|---|---|
| | | NS pH | | NS pI | I | N | S |
| | | # of Ev | rents | # of E | vents | # of E | vents |
| | | (N=x) | x) | (N= | xx) | (N=: | xx) |
| Body System | MedDRA Term | Related n(%) | Not Related n(%) | Related n(%) | Not Related n(%) | Related n(%) | Not Related n(%) |
| Total AEs | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ear and labyrinth disorders | Ear pain | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Total number of subjects in each treatment group in the safety set; n = number of subjects with adverse events in each MedDRA term; Percentages are based on total number of subjects in the safety set within each treatment group

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 04-11pi-2017 |

# T14.1.9.5.13 Summary of Treatment Emergent Adverse Events after 30 Weeks of Study Treatment by Relationship to Study Treatment (Safety Analysis Set) Repeat of T14.1.9.5.12 for after 30 weeks of study treatment

T14.1.9.5.14 Summary of Treatment Emergent Adverse Events of Special Interest by Relationship to Study Treatment (Safety Analysis Set)

Repeat of T14.1.9.5.12 for AESI

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# T14.1.9.5.15 Summary of Treatment Emergent Serious Adverse Events after 52 Weeks of Study Treatment (Safety Analysis Set)

| Body System | MedDRA Term | GSP 301 placebo NS pH (N=xxx) n(%) | GSP 301 placebo<br>NS pH<br>(N=xxx)<br>n(%) | GSP 301<br>NS<br>(N=xxx)<br>n(%) |
|---|---|---|---|---|
| Subject with at least one SAE | Subject with at least one SAE | xxx (xx.x) | xxx(xx.x) | xxx(xx.x) |
| Gastrointestinal disorders | Dry mouth | xxx (xx.x) | xxx (xx.x) | xxx(xx.x) |
| etc. | etc. | | | |

N = Total number of subjects in each treatment group in the safety set;

Percentages are based on total number of subjects in the safety set within each treatment group

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

n = number of subjects with adverse events in each MedDRA term;

|---|---|
| (Study No. GSP 301-303) | r |

### T14.1.9.5.16 Summary of Treatment Emergent Serious Adverse Events after 30 Weeks of Study Treatment (Safety Analysis Set)

Repeat of T14.1.9.5.15 for after 30 weeks of study treatment

### T14.1.9.5.17 Summary of Treatment Related Emergent Serious Adverse Events after 52 Weeks of Study Treatment (Safety Analysis Set)

Repeat of T14.1.9.5.15 for treatment emergent SAE after 52 weeks of study treatment

# T14.1.9.5.18 Summary of Treatment Related Emergent Serious Adverse Events after 30 Weeks of Study Treatment (Safety Analysis Set)

Repeat of T14.1.9.5.15 for treatment emergent SAE after 30 weeks of study treatment

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|
| (Study No. GSP 301-303) | r |

### T14.1.9.5.19.1 Overall Summary of Adverse Events During Placebo Run-In Period (Safety Analysis Set)

| | GSP 301 placebo<br>NS pH | GSP 301 placebo<br>NS pH | GSP 301<br>NS |
|---|---|---|---|
| Subjects in Safety Analysis Set (N1) | XXX | XXX | XXX |
| Subjects with at least one AE n1(%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Discontinued study drug due to above AE n1(%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| AEs reported (N2) | XXX | xxx | xxx |
| Mild n2(%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Moderate n2(%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Severe n2(%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Not Related n2(%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Related n2(%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Death n2(%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Serious AE n2(%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

N2: number of adverse events in treatment group; \$n2(%)\$: percentage based on N2

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

### T14.1.9.5.19.2 Overall Summary of Adverse Events Pre-Randomization

Repeat of T14.1.9.5.19.1 for pre-randomization

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|-------------------------|---------------------|-------------------|
| (Study No. GSP 301-303) | , 4151611 110 | 04-Apr-2017 |

# T14.1.9.6.1 Summary of Clinical laboratory Assessment (Biochemistry) (Safety Analysis Set) Lab Test: xxxxx

| | | _ | Obs | erved Data | | | Change t | from Baseline | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Visit | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pH (N=xxx) | Baseline | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | Visit 8 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | Visit 12 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH (N=xxx) GSP 301 NS (N=xxx)

Baseline is defined as the last available lab values at Screening Visit [Visit 1].

Table will continue for other lab tests.

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 01 11pt 2017 |

T14.1.9.6.2 Summary of Clinical laboratory Assessment (Hematology)
(Safety Analysis Set)
Repeat of T14.1.9.6.1 for hematology

T14.1.9.6.3 Summary of Clinical laboratory Assessment (Urinalysis) (Safety Analysis Set)

Repeat of T14.1.9.6.1 for urinalysis

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### T14.1.9.6.4 Summary of Potentially Clinical Significant Laboratory Results (Biochemistry) (Safety Analysis Set)

Lab Test: xxxxx

| | | Normal | Abnormal | Abnormal (NCS) | Abnormal(CS) |
|---|---|---|---|---|---|
| Treatment Group | Visit | n(%) | n(%) | n(%) | n(%) |
| GSP 301 placebo NS pH (N=xxx) | Baseline | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 8 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 12 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GSP 301 placebo NS pH (N=xxx) GSP 301 NS (N=xxx)

Baseline is defined as the last available lab values at Screening Visit [Visit 1]. CS= Clinically Significant, NCS= Not Clinically Significant

Table will continue for other lab tests.

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 04-11pi-2017 |

T14.1.9.6.5 Summary of Potentially Clinical Significant Laboratory Results (Hematology) (Safety Analysis Set)

Repeat of T14.1.9.6.4 for hematology

T14.1.9.6.6 Summary of Potentially Clinical Significant Laboratory Results (Urinalysis) (Safety Analysis Set)

Repeat of T14.1.9.6.4 for urinalysis

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# T14.1.9.6.7 Shift Tables for Changes from Baseline in Laboratory Results (Biochemistry) to End of Treatment (Safety Analysis Set)

#### Lab Test: xxxxx

| | | End of Treatment | | | |
|---|---|---|---|---|---|
| Treatment Group | Baseline | Normal<br>n (%) | Abnormal n (%) | Abnormal (NCS) n (%) | Abnormal<br>(CS)<br>n (%) |
| GSP 301 placebo NS pH N=xxx) | Normal | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Abnormal | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Abnormal (NCS) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Abnormal (CS) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the last available lab values at Screening Visit [Visit 1]. CS= Clinically Significant, NCS= Not Clinically Significant

Table will continue for other lab tests.

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 04-11pi-2017 |

# T14.1.9.6.8 Shift Tables for Changes from Baseline in Laboratory Results (Hematology) to End of Treatment (Safety Analysis Set)

Repeat of T14.1.9.6.7 for hematology

T14.1.9.6.9 Shift Tables for Changes from Baseline in Laboratory Results (Urinalysis) to End of Treatment (Safety Analysis Set)

Repeat of T14.1.9.6.7 for urinalysis

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| GPL/CT/2014/018/III | 77 ' 10 | SAP Version Date:<br>04-Apr-2017 |
|-------------------------|-------------|----------------------------------|
| (Study No. GSP 301-303) | Version 1.0 | 04-Apr-2017 |

### T14.1.9.7.1 Summary of Vital Signs (Safety Analysis Set)

Systolic Blood Pressure (mmHg)

| | | Observed Data | | | | Change | from Baseline | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Visit | N | Mean (SD) | Median | Min, Max | N | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pH (N=xxx) | Visit 2 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | Visit 8 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | Visit 12 | XX | xx.x (xx.x) | XX.X | xx.x, xx.x | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH (N=xxx)

Baseline is defined as the last available vital signs at Randomization Visit [Visit 2].

Table will continue for Diastolic Blood Pressure (mmHg) and Pulse Rate (bpm).

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

### T14.1.9.7.2 Summary of Potentially Clinical Significant Vital Signs (Safety Analysis Set)

### Systolic Blood Pressure (mmHg)

| | | Normal | Abnormal | Abnormal (NCS) | Abnormal (CS) |
|---|---|---|---|---|---|
| Treatment Group | Visit | n (%) | n (%) | n (%) | n (%) |
| GSP 301 placebo NS pH (N=xxx) | Visit 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 8 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 12 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GSP 301 placebo NS pH (N=xxx) GSP 301 NS (N=xxx)

Baseline is defined as the last available vital signs at Randomization Visit [Visit 2].

CS= Clinically Significant, NCS= Not Clinically Significant

Table will continue for Diastolic Blood Pressure (mmHg) and Pulse Rate (bpm).

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### T14.1.9.7.3 Shift Tables for Changes from Baseline in Vital Signs to End of Treatment (Safety Analysis Set)

### Systolic Blood Pressure (mmHg)

| | | End of Treatment | | | |
|---|---|---|---|---|---|
| | | Normal | Abnormal | Abnormal (NCS) | Abnormal (CS) |
| Treatment Group | Baseline | n (%) | n (%) | n (%) | n (%) |
| GSP 301 placebo NS pH (N=xxx) | Normal | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 1 | Abnormal | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Abnormal (NCS) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Abnormal (CS) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GSP 301 NS (N=xxx)

Baseline is defined as the last available vital signs at Randomization Visit [Visit 2]. CS= Clinically Significant, NCS= Not Clinically Significant

Table will continue for Diastolic Blood Pressure (mmHg) and Pulse Rate (bpm).

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| otocol Number:<br>PL/CT/2014/018/III<br>audy No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|

### T14.1.9.8.1 Summary of ECGs (Safety Analysis Set)

#### PR Interval

| | | | Observed l | Data | | | Change | from Baseline | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Visit | N | Mean (SD) | Median | Min, Max | N | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pH (N=xxx) | Baseline | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | Visit 12 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH (N=xxx) GSP 301 NS (N=xxx)

Baseline is defined as the last available ECG values at Screening Visit [Visit 1].

Table will continue for other ECG parameters.

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III | SAP Version Number:<br>Version 1.0 | SAP Version Date: |
|---|---|---|
| (Study No. GSP 301-303) | Version 1.0 | 04-Apr-2017 |

# T14.1.9.8.2 Summary of Potentially Clinical Significant ECGs (Safety Analysis Set)

| Treatment Group | Visit | Normal<br>n (%) | Abnormal<br>n (%) | Abnormal (NCS)<br>n (%) | Abnormal (CS)<br>n (%) |
|---|---|---|---|---|---|
| GSP 301 placebo NS pH N=xxx) | Baseline | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 12 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the last available ECG values at Screening Visit [Visit 1]. CS= Clinically Significant, NCS= Not Clinically Significant

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

# T14.1.9.8.3 Shift Tables for Changes from Baseline in ECG Interpretation to End of Treatment (Safety Analysis Set)

| | | End of Treatment | | | |
|---|---|---|---|---|---|
| | | Normal | Abnormal | Abnormal (NCS) | Abnormal (CS |
| Treatment Group | Baseline | n (%) | n (%) | n (%) | n (%) |
| GSP 301 placebo NS pH (N=xxx) | Normal | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 1 1 | Abnormal | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Abnormal (NCS) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Abnormal (CS) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the last available ECG values at Screening Visit [Visit 1]. CS= Clinically Significant, NCS= Not Clinically Significant

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|

### T14.1.9.9 Summary of Physical Examinations (Safety Analysis Set)

### **General Appearance**

| | | Normal | Abnormal | Abnormal (NCS) | Abnormal (CS) |
|---|---|---|---|---|---|
| Treatment Group | Visit | n (%) | n (%) | n (%) | n (%) |
| GSP 301 placebo NS pH N=xxx) | Visit 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| • | Visit 8 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 12 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GSP 301 placebo NS pH (N=xxx) GSP 301 NS (N=xxx)

. CS= Clinically Significant, NCS= Not Clinically Significant

Table will continue for other body systems.

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### T14.1.9.10.1 Summary of Focused ENT Examination (Safety Analysis Set)

### **ENT Examination: Nasal Irritation**

| | | | | ENT G | rading | | |
|---|---|---|---|---|---|---|---|
| Γreatment Group | Visit | 0 | 1A | 1B | 2 | 3 | 4 |
| | | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| GSP 301 placebo NS pH<br>N=xxx) | Visit 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 3 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 4 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 5 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 6 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x |
| | Visit 7 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 8 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x |
| | Visit 9 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x |
| | Visit 10 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x |
| | Visit 11 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x |
| | Visit 12 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GSP 301 placebo NS pH N=xxx) GSP 301 NS (N=xxx)

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

### T14.1.9.10.1 Summary of Focused ENT Examination (Safety Analysis Set) (continued)

### **ENT Examination: Epistaxis**

| | ENT Grading | | | | |
|---|---|---|---|---|---|
| Treatment Group | Visit | 0 (None) | 1 (Mild) | 2 (Moderate) | 3 (Severe) |
| | | n (%) | n (%) | n (%) | n (%) |
| | Visit 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| GSP 301 placebo NS pH N=xxx) | Visit 2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 1 | Visit 3 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 4 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 5 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 6 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 7 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 8 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 9 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 10 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 11 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 12 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GSP 301 placebo NS pH (N=xxx) GSP 301 NS (N=xxx)

Programming notes: table will continue for Mucosal Edema , Nasal Discharge , Mucosal Erythema , and Crusting of Mucosa

Data source: xx

 $\label{eq:created on: ddmmmyy hh:mm} Page \ 1 \ of \ N$ 

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|
| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### T14.1.9.10.1 Summary of Focused ENT Examination (Safety Analysis Set) (continued)

#### **ENT Examination:** Throat irritation

| | | ENT | Grading |
|-------------------------------|----------|------------|------------|
| Treatment Group | Visit | Absent | Present |
| | | n (%) | n (%) |
| GSP 301 placebo NS pH (N=xxx) | Visit 1 | xxx (xx.x) | xxx (xx.x) |
| 1 | Visit 2 | xxx (xx.x) | xxx (xx.x) |
| | Visit 3 | xxx (xx.x) | xxx (xx.x) |
| | Visit 4 | xxx (xx.x) | xxx (xx.x) |
| | Visit 5 | xxx (xx.x) | xxx (xx.x) |
| | Visit 6 | xxx (xx.x) | xxx (xx.x) |
| | Visit 7 | xxx (xx.x) | xxx (xx.x) |
| | Visit 8 | xxx (xx.x) | xxx (xx.x) |
| | Visit 9 | xxx (xx.x) | xxx (xx.x) |
| | Visit 10 | xxx (xx.x) | xxx (xx.x) |
| | Visit 11 | xxx (xx.x) | xxx (xx.x) |
| | Visit 12 | xxx (xx.x) | xxx (xx.x) |

GSP 301 placebo NS pH (N=xxx) GSP 301 NS (N=xxx)

Programming notes: table will continue for candidiasis, post nasal drip.

Data source: xx

|---|---|---|

T14.1.9.10.2 Summary of Potentially Clinical Significant Focused ENT Examination (Safety Analysis Set)

#### Nasal Irritation

| | | Normal | Abnormal | Abnormal (NCS) | Abnormal (CS) |
|---|---|---|---|---|---|
| Treatment Group | Visit | n(%) | n(%) | n(%) | n(%) |
| | Visit 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| GSP 301 placebo NS pH (N=xxx) | Visit 2 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 1 | Visit 3 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 4 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 5 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 6 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 7 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 8 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 9 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 10 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 11 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | Visit 12 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

GSP 301 placebo NS pH (N=xxx) GSP 301 NS (N=xxx)

Table will continue for other evaluations.

<sup>.</sup> CS= Clinically Significant, NCS= Not Clinically Significant

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

T14.1.9.11.1 Summary of Extent of Exposure during the Post Randomization Treatment Period (Safety Analysis Set)

| | | GSP 301 placebo | GSP 301 placebo | GSP 301 |
|---|---|---|---|---|
| | | NS pĤ | NS pH | NS |
| | | (N=xxx) | (N=xxx) | (N=xxx) |
| Number of days on treatment | n | XXX | XXX | XXX |
| | Mean $\pm$ SD | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x |
| Number of days on study | n | xxx | xxx | xxx |
| • | Mean $\pm$ SD | $xx.x \pm x.x$ | $xx.x \pm x.x$ | $xx.x \pm x.x$ |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Treatment Compliance n (%) | <75% | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 1 | >=75% - <=100% | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | >100% - =<125% | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | >125% | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

N= number of subjects in the treatment group; n= number of subject with data available;

Number of days on study = End of Study Date - Enrollment Date (Screening Visit) +1

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 04-11pi-2017 |

# T14.1.9.11.2 Summary of Rescue Medication (Safety Analysis Set)

| Rescue medication | GSP 301 placebo | GSP 301 placebo | GSP 301 |
|-------------------|-----------------|-----------------|------------|
| | NS pH | NS pH | NS |
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Loratadine n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| etc | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| etc | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

N= number of subjects in the treatment group; n= number of subject with data available;

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | 77 . 10 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### T14.1.9.12.1 Summary of Average AM rTNSS (Full Analysis Set)

| | | | Obs | erved Data | | _ | Chang | e from Baseline | e |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Week | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pH (N=xxx) | Baseline | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | 1 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | 2 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x(xx.x) | XX.X | XX.X, XX.X |
| | etc | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x(xx.x) | XX.X | XX.X, XX.X |
| | 52 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the mean of the last 4 AM reading scores including the AM on the day of randomization

Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available;

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

### T14.1.9.12.2 Summary of Repeated Measures Analysis Results in Average AM rTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)

| | | | | | Tre | eatment vs. Plac | ebo NS pH | |
|---|---|---|---|---|---|---|---|---|
| Week | Treatment | Number of | I CM | Std Err | LSMean | Std Err | 059/ GI | D 1 |
| | Group | Subjects (n) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| 6 Weeks | GSP 301 placebo NS pH (N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| 30 Weeks | GSP 301 placebo NS pH N=xxx) | xxx | xxx.xx | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | x.xxxx |
| 52 Weeks | GSP 301 placebo NS pH (N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.x - xx.x | X.XXXX |

Baseline is defined as the mean of the last 4 AM reading scores including the AM on the day of randomization

LSMeans: Least square means; Std Err LSMeans: Standard error of the LSMeans

LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on separate mixed model repeated measures models for each week assessment, with change from baseline as dependent variable, treatment group and site as fixed effect, baseline as covariate, and week as the within-subject effect.

Programming note: the interaction terms treatment\*baseline and treatment\*site will only be included in the footnote if significant in the model

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

n: Number of subjects with data available in the specific treatment group

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### T14.1.9.12.3 Summary of Average AM rTNSS (Per Protocol Set)

Repeat of Table T14.1.9.12.1 for Per Protocol Set

#### T14.1.9.12.4 Summary of Repeated Measures Analysis Results in Average AM rTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set)

Repeat of Table T14.1.9.12.2 for Per Protocol Set

### T14.1.9.12.5 Subgroup Analyses (Age Group): Summary of Average AM rTNSS (Full Analysis Set) Repeat of Table T14.1.9.12.1 for age group

### T14.1.9.12.6 Subgroup Analyses (Sex): Summary of Average AM rTNSS (Full Analysis Set)

Repeat of Table T14.1.9.12.1 for sex

### T14.1.9.12.7 Subgroup Analyses (Race): Summary of Average AM rTNSS (Full Analysis Set)

Repeat of Table T14.1.9.12.1 for race

#### T14.1.9.12.8 Subgroup Analyses (Ethnicity): Summary of Average AM rTNSS (Full Analysis Set)

Repeat of Table T14.1.9.12.1 for ethnicity

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

# T14.1.9.13.1 Summary of Average AM iTNSS (Full Analysis Set)

| | | | Obs | erved Data | | _ | Chang | e from Baseline | 2 |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Week | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pH (N=xxx) | Baseline | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | 1 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | 2 | XX | xx.x(xx.x) | XX.X | XX.X, XX.X | XX | xx.x(xx.x) | XX.X | XX.X, XX.X |
| | etc | XX | xx.x(xx.x) | XX.X | XX.X, XX.X | XX | xx.x(xx.x) | XX.X | XX.X, XX.X |
| | 52 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x(xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the mean of the last 4 AM reading scores including the AM on the day of randomization

Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available;

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### T14.1.9.13.2 Summary of Repeated Measures Analysis Results in Average AM iTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)

| | | | | | Tre | eatment vs. Plac | ebo NS pH | |
|---|---|---|---|---|---|---|---|---|
| Week | Treatment | Number of | | Std Err | LSMean | Std Err | <u> </u> | |
| | Group | Subjects (n) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| 6 Weeks | GSP 301 placebo NS pH N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| 30 Weeks | GSP 301 placebo NS pH (N=xxx) | xxx | xxx.xx | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| 52 Weeks | GSP 301 placebo NS pH N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.x - xx.x | X.XXXX |

Baseline is defined as the mean of the last 4 AM reading scores including the AM on the day of randomization

LSMeans: Least square means; Std Err LSMeans: Standard error of the LSMeans

LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on separate mixed model repeated measures models for each week assessment, with change from baseline as dependent variable, treatment group and site as fixed effect, baseline as covariate, and week as the within-subject effect.

Programming note: the interaction terms treatment\*baseline and treatment\*site will only be included in the footnote if significant in the model

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

n: Number of subjects with data available in the specific treatment group

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# T14.1.9.13.3 Summary of Average AM iTNSS (Per Protocol Set)

Repeat of Table T14.1.9.13.1 for Per Protocol Set

#### T14.1.9.13.4 Summary of Repeated Measures Analysis Results in Average AM iTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set)

Repeat of Table T14.1.9.13.2 for Per Protocol Set

## T14.1.9.13.5 Subgroup Analyses (Age Group): Summary of Average AM iTNSS (Full Analysis Set)

Repeat of Table T14.1.9.13.1 for age group

### T14.1.9.13.6 Subgroup Analyses (Sex): Summary of Average AM iTNSS (Full Analysis Set) Repeat of Table T14.1.9.13.1 for sex

### T14.1.9.13.7 Subgroup Analyses (Race): Summary of Average AM iTNSS (Full Analysis Set)

Repeat of Table T14.1.9.13.1 for race

#### T14.1.9.13.8 Subgroup Analyses (Ethnicity): Summary of Average AM iTNSS (Full Analysis Set)

Repeat of Table T14.1.9.13.1 for ethnicity

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

# T14.1.9.14.1 Summary of the Overall RQLQ(S) (Full Analysis Set)

| | | | Obs | erved Data | | | Chang | e from Baselin | e |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Week | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pH N=xxx) | Baseline | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | 6 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | 30 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | 52 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the RQLQ(S) score at the randomization visit.

Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available;

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### T14.1.9.14.2 Summary of Repeated Measures Analysis Results in Overall RQLQ(S) at Weeks 6, 30, and 52 (Full Analysis Set)

| | | | | | Tre | eatment vs. Plac | ebo NS pH | |
|---|---|---|---|---|---|---|---|---|
| Week | Treatment | Number of | | Std Err | LSMean | Std Err | | |
| | Group | Subjects (n) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| Week 6 | GSP 301 placebo NS pH (N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| Week 30 | GSP 301 placebo NS pH N=xxx) | xxx | xxx.xx | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| Week 52 | GSP 301 placebo NS pF | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX,XX | XXX.XX | XXX,XX | xx.x - xx.x | X.XXXX |

Baseline is defined as the RQLQ(S) score at the randomization visit.

LSMeans: Least square means; Std Err LSMeans: Standard error of the LSMeans

LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on mixed model repeated measures model with change from baseline as dependent variable, treatment group and site as fixed effect, baseline as covariate, week as the within-subject effect and week-by-treatment interaction.

Programming note: the interaction terms treatment\*baseline and treatment\*site will only be included in the footnote if significant in the model

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

n: Number of subjects with data available in the specific treatment group

| D ( 131 1 | CADA : N. 1 | |
|-------------------------|---------------------|-------------------|
| (Study No. GSP 301-303) | | 04-Apr-2017 |

# T14.1.9.14.3 Summary of Overall RQLQ(S) (RQLQ(S) Analysis Set) Repeat of Table T14.1.9.14.1 for RQLQ(S) Analysis Set

T14.1.9.14.4 Summary of Repeated Measures Analysis Results in Overall RQLQ(S) at Weeks 6, 30, and 52 (RQLQ(S) Analysis Set)

Repeat of Table T14.1.9.14.2 for RQLQ(S) Analysis Set

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

### T14.1.9.15.1 Summary of Average AM Reflective Individual Nasal Symptoms (Full Analysis Set) Rhinorrhea

| | | | | ixiiiiioi i iica | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Obs | erved Data | | | Chang | e from Baseline | e |
| Treatment Group | Week | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pF (N=xxx) | Baseline | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | 1 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | 2 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | etc | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | 52 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the mean of the last 4 AM reading scores including the AM on the day of randomization

Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available;

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Programming notes: table will continue for other nasal symptom scores (nasal congestion, nasal itching, and sneezing).

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# T14.1.9.15.2 Summary of Repeated Measures Analysis Results in Average AM Reflective Individual Nasal Symptoms over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)

### Rhinorrhea

| | | | | | Tre | eatment vs. Plac | ebo NS pH | |
|---|---|---|---|---|---|---|---|---|
| Week | Treatment | Number of | | Std Err | LSMean | Std Err | | |
| | Group | Subjects (n) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| 6 Weeks | GSP 301 placebo NS pH N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | xxx.xx | XXX.XX | XXX.XX | xx.xx - xx.xx | x.xxxx |
| 30 Weeks | GSP 301 placebo NS pH (N=xxx) | xxx | xxx.xx | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| 52 Weeks | GSP 301 placebo NS pH (N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.x - xx.x | X.XXXX |

Baseline is defined as the mean of the last 4 AM reading scores including the AM on the day of randomization

LSMeans: Least square means; Std Err LSMeans: Standard error of the LSMeans

LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on separate mixed model repeated measures models for each week assessment, with change from baseline as dependent variable, treatment group and site as fixed effect, baseline as covariate, and week as the within-subject effect.

Programming note: the interaction terms treatment\*baseline and treatment\*site will only be included in the footnote if significant in the model Programming notes: table will continue for other nasal symptom scores (nasal congestion, nasal itching, and sneezing).

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

n: Number of subjects with data available in the specific treatment group

| D ( 131 1 | CADA : N. 1 | |
|-------------------------|---------------------|-------------------|
| (Study No. GSP 301-303) | | 04-Apr-2017 |

# T14.1.9.16.1 Summary of Average AM Instantaneous Individual Nasal Symptoms (Full Analysis Set) Repeat of Table T14.1.9.15.1 for Instantaneous Individual Nasal Symptoms

T14.1.9.16.2 Summary of Repeated Measures Analysis Results in Average AM Instantaneous Individual Nasal Symptoms over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)

Repeat of Table T14.1.9.15.2 for Instantaneous Individual Nasal Symptoms

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### T14.1.9.17.1 Summary of Repeated Measures Analysis Results in Average AM rTNSS over Each Treatment Week (Full Analysis Set)

| | | | | | Tre | eatment vs. Plac | ebo NS pH | |
|---|---|---|---|---|---|---|---|---|
| Week | Treatment | Number of | | Std Err | LSMean | Std Err | | |
| | Group | Subjects (n) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| Week 1 | GSP 301 placebo NS pH (N=xxx) | xxx | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | xxx.xx | xxx.xx | XXX.XX | XXX.XX | xx.xx - xx.xx | x.xxxx |
| etc | GSP 301 placebo NS pH N=xxx) | xxx | xxx.xx | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| Week 52 | GSP 301 placebo NS pH | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.x - xx.x | X.XXXX |

Baseline is defined as the mean of the last 4 AM reading scores including the AM on the day of randomization

LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on mixed model repeated measures model with change from baseline as dependent variable, treatment group and site as fixed effect, baseline as covariate, week as the within-subject effect and week-by-treatment interaction.

Programming note: the interaction terms treatment\*baseline and treatment\*site will only be included in the footnote if significant in the model

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

n: Number of subjects with data available in the specific treatment group

 $LSMeans: Least \ square \ means; \ \ Std \ Err \ LSMeans: Standard \ error \ of \ the \ LSMeans$ 

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 04-11pi-2017 |

T14.1.9.17.2 Summary of Repeated Measures Analysis Results in Average AM iTNSS over Each Treatment Week (Full Analysis Set)

Repeat of Table T14.1.9.17.1 for iTNSS

|---|---|
| (Study No. GSP 301-303) | r |

### T14.1.9.18.1 Summary of Repeated Measures Analysis Results in Average AM Subject-reported Reflective Individual Nasal Symptoms over Each Treatment Week

### (Full Analysis Set)

### Rhinorrhea

| | | | | | Tre | eatment vs. Plac | ebo NS pH | |
|---|---|---|---|---|---|---|---|---|
| Week | Treatment | Number of | | Std Err | LSMean | Std Err | | |
| | Group | Subjects (n) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| Week 1 | GSP 301 placebo NS pH (N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| etc | GSP 301 placebo NS pH (N=xxx) | xxx | xxx.xx | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | x.xxxx |
| Week 52 | GSP 301 placebo NS pH (N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.x - xx.x | X.XXXX |

Baseline is defined as the mean of the last 4 AM reading scores including the AM on the day of randomization

LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on mixed model repeated measures model with change from baseline as dependent variable, treatment group and site as fixed effect, baseline as covariate, week as the within-subject effect and week-by-treatment interaction.

Programming note: the interaction terms treatment\*baseline and treatment\*site will only be included in the footnote if significant in the model Programming notes: table will continue for other nasal symptom scores (nasal congestion, nasal itching, and sneezing).

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

n: Number of subjects with data available in the specific treatment group

LSMeans: Least square means; Std Err LSMeans: Standard error of the LSMeans

| ſ | D . 137 1 | GADAY : N. 1 | |
|---|---|---|---|
| | (Study No. GSP 301-303) | , | 04-Api-201/ |

T14.1.9.18.2 Summary of Repeated Measures Analysis Results in Average AM Subject-reported Instantaneous Individual
Nasal Symptoms over Each Treatment Week
(Full Analysis Set)
Repeat of Table T14.1.9.18.1 for instantaneous individual nasal symptoms

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

# T14.1.9.19.1 Summary of the Physician Assessed Nasal Symptom Score (PNSS) (Full Analysis Set)

| | | | Obs | erved Data | | _ | Chang | e from Baselin | e |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Week | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pF (N=xxx) | Baseline | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | 3 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | etc | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x(xx.x) | XX.X | XX.X, XX.X |
| | 52 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the PNSS score at the randomization visit.

Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available;

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

### T14.1.9.19.2 Summary of Repeated Measures Analysis Results in Physician Assessed Nasal Symptom Score (PNSS) at Weeks 6, 30, and 52 (Full Analysis Set)

| | | | | | Tre | eatment vs. Plac | ebo NS pH | |
|---|---|---|---|---|---|---|---|---|
| Week | Treatment | Number of | | Std Err | LSMean | Std Err | | |
| | Group | Subjects (n) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| Week 6 | GSP 301 placebo NS pH (N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| Week 30 | GSP 301 placebo NS pH (N=xxx) | xxx | xxx.xx | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| Week 52 | GSP 301 placebo NS pH N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.x - xx.x | X.XXXX |

Baseline is defined as the PNSS score at the randomization visit.

n: Number of subjects with data available in the specific treatment group

LSMeans: Least square means; Std Err LSMeans: Standard error of the LSMeans

LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on mixed model repeated measures model with change from baseline as dependent variable, treatment group and site as fixed effect, baseline as covariate, week as the within-subject effect and week-by-treatment interaction.

Programming note: the interaction terms treatment\*baseline and treatment\*site will only be included in the footnote if significant in the model

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

# T14.1.9.20.1 Summary of the Physician Assessed Individual Nasal Symptom Score (Full Analysis Set)

**Runny Nose** 

| | | _ | Obs | erved Data | | _ | Chang | e from Baseline | e |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Week | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pH (N=xxx) | Baseline | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | 3 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | etc | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x(xx.x) | XX.X | XX.X, XX.X |
| | 52 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the nasal symptom score at the randomization visit.

Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available;

Data source: xx

Created on: ddmmmyy hh:mm  $\qquad \qquad \text{Page 1 of N}$ 

Programming notes: table will continue for other nasal symptom scores (nasal congestion, nasal itching, and sneezing).

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

## T14.1.9.20.2 Summary of Repeated Measures Analysis Results in Physician Assessed Individual Nasal Symptom Score at Weeks 6, 30, and 52 (Full Analysis Set)

| | Running Nose | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | Tre | ebo NS pH | | |
| Week | Treatment | Number of | | Std Err | LSMean | Std Err | | |
| | Group | Subjects (n) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| Week 6 | GSP 301 placebo NS pF | XXX | XXX.XX | XXX.XX | | | | _ |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | xxx.xx | XXX.XX | xxx.xx | xx.xx - xx.xx | x.xxxx |
| Week 30 | GSP 301 placebo NS pH N=xxx) | xxx | xxx.xx | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| Week 52 | GSP 301 placebo NS pH (N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.x - xx.x | X.XXXX |

Baseline is defined as the nasal symptom score at the randomization visit.

LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on mixed model repeated measures model with change from baseline as dependent variable, treatment group and site as fixed effect, baseline as covariate, week as the within-subject effect and week-by-treatment interaction.

Programming note: the interaction terms treatment\*baseline and treatment\*site will only be included in the footnote if significant in the model Programming notes: table will continue for other nasal symptom scores (nasal congestion, nasal itching, and sneezing).

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

n: Number of subjects with data available in the specific treatment group

LSMeans: Least square means; Std Err LSMeans: Standard error of the LSMeans

|---|---|---|

### T14.1.9.21.1 Summary of the Individual Domains of the RQLQ(S) (Full Analysis Set)

#### Emotional

| | | | | Linotionai | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Obs | erved Data | | | Change | e from Baseline | ē |
| Treatment Group | Week | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pH N=xxx) | Baseline | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | 3 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | etc | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | 52 | XX | xx.x(xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the domain score at the randomization visit.

Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available;

Data source: xx

Programming notes: table will continue for other domains.

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### T14.1.9.21.2 Summary of Repeated Measures Analysis Results in the Individual Domains of the RQLQ(S) at Weeks 6, 30, and 52 (Full Analysis Set)

#### **Emotional**

| | | | | | Tre | eatment vs. Plac | ebo NS pH | |
|---|---|---|---|---|---|---|---|---|
| Week | Treatment | Number of | | Std Err | LSMean | Std Err | | |
| | Group | Subjects (n) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| Week 6 | GSP 301 placebo NS pH (N=xxx) | XXX | XXX.XX | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | x.xxxx |
| Week 30 | GSP 301 placebo NS pH (N=xxx) | xxx | xxx.xx | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| Week 52 | GSP 301 placebo NS pH | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.x - xx.x | X.XXXX |

Baseline is defined as the domain score at the randomization visit.

LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on mixed model repeated measures model with change from baseline as dependent variable, treatment group and site as fixed effect, baseline as covariate, week as the within-subject effect and week-by-treatment interaction.

Programming note: the interaction terms treatment\*baseline and treatment\*site will only be included in the footnote if significant in the model Programming notes: table will continue for other domains

Data source: xx

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

n: Number of subjects with data available in the specific treatment group

LSMeans: Least square means; Std Err LSMeans: Standard error of the LSMeans

|-------------------------|---------------------|-------------------|
| (Study No. GSP 301-303) | , Gibion 1.0 | 04-Apr-2017 |

# T14.1.9.21.3 Summary of the Individual Domains of the RQLQ(S) (RQLQ(S) Analysis Set) Repeat of Table T14.1.9.21.1 for RQLQ(S) Analysis Set

T14.1.9.21.4 Summary of Repeated Measures Analysis Results in the Individual Domains of the RQLQ(S) at Weeks 6, 30, and 52 (RQLQ(S) Analysis Set)

Repeat of Table T14.1.9.21.2 for RQLQ(S) Analysis Set

|--------------------------|--------------|----------------|
|--------------------------|--------------|----------------|

|---|---|---|

# T14.1.9.22.1 Summary of RCAT (Full Analysis Set)

| | | _ | Observed Data | | | | Change from Baseline | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Week | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pH (N=xxx) | Baseline | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | 3 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | etc | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | 52 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the RCAT score at the randomization visit.

Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available;

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Programming notes: table will continue for other domains.

|--------------------------|--------------|-----------------|
|--------------------------|--------------|-----------------|

|---|---|---|

# T14.1.9.22.2 Summary of Repeated Measures Analysis Results in RCAT at Weeks 6, 30, and 52 (Full Analysis Set) Domain 1

| | | | Doman | 1 1 | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | Tre | İ | | |
| Week | Treatment | Number of | | Std Err | LSMean | Std Err | | |
| | Group | Subjects (n) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| Week 6 | GSP 301 placebo NS pH (N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | xxx.xx | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | x.xxxx |
| Week 30 | GSP 301 placebo NS pH (N=xxx) | xxx | xxx.xx | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| Week 52 | GSP 301 placebo NS pH | XXX | xxx.xx | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.x - xx.x | X.XXXX |

Baseline is defined as the RCAT score at the randomization visit.

LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on mixed model repeated measures model with change from baseline as dependent variable, treatment group and site as fixed effect, baseline as covariate, week as the within-subject effect and week-by-treatment interaction.

Programming note: the interaction terms treatment\*baseline and treatment\*site will only be included in the footnote if significant in the model Programming notes: table will continue for other domains

Data source: xx

|--------------------------|--------------|-----------------|
|--------------------------|--------------|-----------------|

n: Number of subjects with data available in the specific treatment group

LSMeans: Least square means; Std Err LSMeans: Standard error of the LSMeans

|---|---|---|

### T14.1.9.23.1 Summary of the Individual Domains of the RCAT (Full Analysis Set)

#### Domain 1

| | | | | Domain 1 | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | _ | Obs | erved Data | | | Chang | e from Baseline | <u>.</u> |
| Treatment Group | Week | n | Mean (SD) | Median | Min, Max | n | Mean (SD) | Median | Min, Max |
| GSP 301 placebo NS pH (N=xxx) | Baseline | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | | | | |
| | 3 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | etc | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |
| | 52 | XX | xx.x (xx.x) | XX.X | XX.X, XX.X | XX | xx.x (xx.x) | XX.X | XX.X, XX.X |

GSP 301 placebo NS pH GSP 301 NS (N=xxx)

Baseline is defined as the domain score at the randomization visit.

Max=maximum; Min=minimum; N= number of subjects in the treatment group; n= number of subjects with data available;

Data source: xx

Programming notes: table will continue for other domains.

|--------------------------|--------------|-----------------|
|--------------------------|--------------|-----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# T14.1.9.23.2 Summary of Repeated Measures Analysis Results in the Individual Domains of the RCAT at Weeks 6, 30, and 52 (Full Analysis Set) Domain 1

| | | | Doman | * * | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | Treatment vs. Placebo NS pH | | | |
| Week | Treatment | Number of | | Std Err | LSMean | Std Err | | |
| | Group | Subjects (n) | LSMean | LSMean | Difference | Difference | 95% CI | P-value |
| Week 6 | GSP 301 placebo NS pH N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| Week 30 | GSP 301 placebo NS pH (N=xxx) | xxx | xxx.xx | xxx.xx | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX.XX | XXX.XX | XXX.XX | XXX.XX | xx.xx - xx.xx | X.XXXX |
| Week 52 | GSP 301 placebo NS pH (N=xxx) | XXX | XXX.XX | XXX.XX | | | | |
| | GSP 301 NS (N=xxx) | XXX | XXX,XX | XXX.XX | XXX.XX | XXX.XX | xx.x - xx.x | X.XXXX |

Baseline is defined as the domain score at the randomization visit.

LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on mixed model repeated measures model with change from baseline as dependent variable, treatment group and site as fixed effect, baseline as covariate, week as the within-subject effect and week-by-treatment interaction.

Programming note: the interaction terms treatment\*baseline and treatment\*site will only be included in the footnote if significant in the model Programming notes: table will continue for other domains

Data source: xx

|--------------------------|--------------|-----------------|
|--------------------------|--------------|-----------------|

n: Number of subjects with data available in the specific treatment group

LSMeans: Least square means; Std Err LSMeans: Standard error of the LSMeans

|-------------------------|---------------------|-------------------|
| (Study No. GSP 301-303) | V 6151611 11.0 | 04-Apr-2017 |

### L16.2.1 Listing of Subject Disposition (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Date of<br>Last Dose<br>Taken | Date of Completion/<br>Early Termination/<br>Withdrawal | Reason for<br>Early Termination/<br>Withdrawal |
|---|---|---|---|---|
| GSP 301 placebo NS pH | xx-xxx/xxxxx | ddmmmyyyy | ddmmmyyyy | Adverse Event |

GSP 301 placebo NS pH GSP 301 NS

Data source: xx

Created on: ddmmmyy hh:mm


|--------------------------|--------------|-----------------|
|--------------------------|--------------|-----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | 77 . 10 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|

### L16.2.2 Listing of Protocol Deviations (Safety Analysis Set)

| Subject /<br>Randomization<br>Number | Deviation Occurred<br>During | Event Description |
|---|---|---|
| xx-xxx/xxxxx | Randomized Treatment | Outside Visit Window (Visit # 4) |
| • | | |
| | Randomization<br>Number | Randomization Deviation Occurred<br>Number During |

Data source: xx

|--------------------------|--------------|-----------------|
|--------------------------|--------------|-----------------|

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### L16.2.3.1 Listing of Subject Excluded from the Per Protocol Set

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Exclusion Reason |
|---|---|---|
| GSP 301 placebo NS pH | xx-xxx/xxxxx | Subject did not meet IE criterion |
| GSP 301 placebo NS pH<br>GSP 301 NS | | |
| Data source: xx<br>Created on: ddmmmyy hh:mm | Page I of N | |

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 04-Api-201/ |

### L16.2.3.2 Listing of Subject Excluded from the Full Analysis Set

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Exclusion Reason |
|---|---|---|
| GSP 301 placebo NS pH | xx-xxx/xxxxx | Subject did not have at least one post- randomization evaluation |
| GSP 301 placebo NS pH<br>GSP 301 NS | | |
| Data source: xx<br>Created on: ddmmmyy hh:mm | Page 1 of N | |

|--------------------------|--------------|-----------------|

|-------------------------|-----------------------|-------------------|
| (Study No. GSP 301-303) | , <b>41</b> 01011 1.0 | 04-Apr-201/ |

### L16.2.3.3 Listing of Subjects Who Withdrew Due to Inclusion/Exclusion Criteria (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Inclusion/Exclusion Criteria |
|---|---|---|
| GSP 301 placebo NS pH | xx-xxx/xxxxx | Exclusion Criteria #1: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| GSP 301 placebo NS pH<br>GSP 301 NS | | |
| ata source: xx | | |

Page 1 of N Created on: ddmmmyy hh:mm

|--------------------------|--------------|-----------------|
|-------------------------|---------------------|-------------------|--|
| (Study No. GSP 301-303) | V GIBIOII 1.0 | 04-Api-201/ | |

#### L16.2.4.1 Listing of Demographic Data (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Age | Sex | Ethnicity | Race | Weight (kg) |
|---|---|---|---|---|---|---|
| GSP 301 placebo NS pH | xx-xxx/xxxxx | 42 | Male | Hispanic or Latino | Black/ African American | XX.X |
| • | xx-xxx/xxxxx | 35 | Female | Hispanic or Latino | White | |
| GSP 301 placebo NS pH<br>GSP 301 NS | | | | | | |

Data source: xx

Created on: ddmmmyy hh:mm


|--------------------------|--------------|-----------------|
|--------------------------|--------------|-----------------|

|-------------------------|-----------------------|-------------------|
| (Study No. GSP 301-303) | , <b>6</b> 101011 1.0 | 04-Apr-201/ |

#### L16.2.4.2 Listing of Medical History (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Body System | Condition/Procedure | Start Date/<br>End Date | Ongoing | Severity<br>Grade | Any Nasal<br>Structural<br>Abnormalities? |
|---|---|---|---|---|---|---|---|
| GSP 301 placebo NS<br>pH | xx-xxx/xxxxx | Respiratory System | xxxxxxxxxxxx | ddmmmyyyy/<br>ddmmmyyyy | No | Mild | No |
| , | xx-xxx/xxxxx | Cardiovascular<br>System | xxxxxxxxxxx | ddmmmyyyy/ | Yes | | Yes (xxxx) |

GSP 301 placebo NS pH GSP 301 NS

Data source: xx

Created on: ddmmmyy hh:mm  $Page \ 1 \ of \ N$ 

|--------------------------|--------------|-----------------|
|--------------------------|--------------|-----------------|

|---|---|
| (Study No. GSP 301-303) | r |

# L16.2.4.3 Listing of Concomitant Medication (Safety Analysis Set)

| Treatment Group | Subject /<br>Randomization<br>Number | Type of<br>Medication | Medication<br>Name | Dose | Frequency | Route | Start Date/<br>End Date | Indication |
|---|---|---|---|---|---|---|---|---|
| GSP 301 placebo<br>NS pH | xx-xxx/xxxxx | Prior | xxxxxxxxxxx | 20mg | QD | PO | ddmmmyyyy/<br>ddmmmyyyy | xxxxxxxxxx |
| 149 h11 | xx-xxx/xxxxx | Concomitant | xxxxxxxxxxx | 10mg | QD | PO | ddmmmyyyy/ | xxxxxxxxxx |

GSP 301 placebo NS pH GSP 301 NS

Data source: xx

Created on: ddmmmyy hh:mm


L16.2.4.4 Listing of Rescue Medication (Safety Analysis Set)

Repeat of Listing L16.2.4.3 for rescue medication

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# L16.2.4.5 Listing of Skin Test and Wheal Measurements (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Test<br>Date | Allergen | Wheal<br>Diameter<br>(mm) | PAR-inducing<br>allergen 3 mm<br>greater than the<br>negative control? | Expected to be exposed to the above specified PAR allergen? |
|---|---|---|---|---|---|---|
| GSP 301 placebo NS pH | xx-xxx/xxxxx | ddmmmyyyy | XXX | XXX | XXX | Yes |

GSP 301 placebo NS pH GSP 301 NS

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 011pr 2017 |

# L16.2.5.1 Listing of Visit Date Information (Safety Analysis Set)

| | Subject / | Informed | | | | | | Visit 11/ |
|---|---|---|---|---|---|---|---|---|
| Treatment | Randomization | Consent | Visit 1/ | Visit 3/ | Visit 5/ | Visit 7/ | Visit 9/ | Visit 12/ |
| Group | Number | Date | Visit 2 | Visit 4 | Visit 6 | Visit 8 | Visit 10 | Early termination |
| GSP 301 | xx-xxx/xxxxx | ddmmmyyyy | ddmmmyyyy/ | ddmmmyyyy/ | ddmmmyyyy/ | ddmmmyyyy/ | ddmmmyyyy/ | ddmmmyyyy/ |
| placebo NS | | 2222 | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy |
| рН | | | | ,,,,,, | | | | |

GSP 301 placebo NS pH GSP 301 NS

Data source: xx

Created on: ddmmmyy hh:mm


Glenmark 

|---|---|---|

#### L16.2.5.2 Listing of Study Compliance (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Visit | Was the used study medication collected? | Was Diary 2 collected and reviewed? | Date of last<br>entry in Diary<br>2 | Total number<br>of confirmed<br>doses applied<br>in Diary 2 | Wa the subject<br>retrained on<br>proper use of<br>the nasal<br>spray? | Was the<br>study<br>medication<br>primed and<br>dispensed? | Was the AR assessment Diary 3 distributed? |
|---|---|---|---|---|---|---|---|---|---|
| GSP 301<br>placebo NS<br>pH | xx-xxx/xxxxx | Visit 3 | Yes | Yes | ddmmmyyyy | xx | Yes | Yes | Yes |
| | | Visit 8<br>Visit 12 | Yes<br>Yes | Yes<br>Yes | ddmmmyyyy<br>ddmmmyyyy | xx<br>xx | Yes<br>Yes | Yes<br>Yes | Yes<br>Yes |

GSP 301 placebo NS pH GSP 301 NS

Data source: xx

Created on: ddmmmyy hh:mm


Glenmark 

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 011pr 2017 |

#### L16.2.5.3 Listing of Extent of Exposure (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Date of<br>First Dose<br>Taken | Date of<br>Last Dose<br>Taken | Number of<br>Days on<br>Treatment | Date of<br>Inform<br>Consent<br>Date | Date of<br>Completion/<br>Early Termination/<br>Withdrawal | Number of<br>Days on<br>Study |
|---|---|---|---|---|---|---|---|
| GSP 301 placebo NS pH | xx-xxx/xxxxx | ddmmmyyyy | ddmmmyyyy | XXX | ddmmmyyyy | ddmmmyyyy | XXX |

GSP 301 placebo NS pH GSP 301 NS

Data source: xx

Created on: ddmmmyy hh:mm


Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# L16.2.6.1 Listing of AM Reflective Nasal Symptom Scores (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Day/Week | Date | Dosing<br>Time | Assessment<br>Time | Rhinorrhea | Nasal<br>Congestion | Nasal<br>Itching | Sneezing | rTNSS |
|---|---|---|---|---|---|---|---|---|---|---|
| GSP 301 placebo<br>NS pH | xx-xxx/xxxxx | Day -7 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| 1 | | Day -6 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | Day -5 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | etc | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | Day -1 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | Day 1/Week 1 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | Week 3 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | etc | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | Week 52 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |

GSP 301 placebo NS pH GSP 301 NS

rTNSS = sum of four nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing)

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

#### L16.2.6.2 Listing of AM Instantaneous Nasal Symptom Scores (Safety Analysis Set)

| T | Subject / | | | Daning | A | | N1 | N1 | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Randomization | | | Dosing | Assessment | | Nasal | Nasal | | |
| Group | Number | Day/Week | Date | Time | Time | Rhinorrhea | Congestion | Itching | Sneezing | rTNSS |
| GSP 301 placebo<br>NS pH | xx-xxx/xxxxx | Day -7 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| 1 | | Day -6 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | Day -5 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | etc | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | Day -1 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | Day 1/Week 1 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | Week 3 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | etc | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |
| | | Week 52 | ddmmmyyy | hh:mm | hh:mm | 0 | 0 | 1 | 0 | 1 |

GSP 301 placebo NS pH GSP 301 NS

iTNSS = sum of four nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing)

Data source: xx

Glenmark 

|---|---|---|

### L16.2.6.3 Listing of the Average AM Reflective Nasal Symptom Scores (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Week | Rhinorrhea | Nasal<br>Congestion | Nasal<br>Itching | Sneezing | rTNSS |
|---|---|---|---|---|---|---|---|
| GSP 301 placebo | xx-xxx/xxxxx | Baseline | XX | xx | XX | xx | XX |
| NS pH | | | | | | | |
| 1 | | Week 1 | XX | XX | XX | XX | XX |
| | | Week 2 | XX | XX | XX | XX | XX |
| | | Week 3 | XX | XX | XX | XX | XX |
| | | Week 4 | XX | XX | XX | XX | XX |
| | | Week 5 | XX | XX | XX | XX | XX |
| | | Week 6 | XX | XX | XX | XX | XX |
| | | etc | XX | XX | XX | XX | XX |
| | | Week 30 | XX | XX | XX | XX | XX |
| | | etc | XX | XX | XX | XX | XX |
| | | Week 52 | XX | XX | XX | XX | XX |

GSP 301 placebo NS pH GSP 301 NS

rTNSS = sum of four nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing)

Baseline is defined as the average of the last 4 consecutive AM assessments during the last 4 days of the run-in period from the Day -3 AM assessment to the AM assessment on the day of randomization.

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# L16.2.6.4 Listing of the Average AM Instantaneous Nasal Symptom Scores (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Week | Rhinorrhea | Nasal<br>Congestion | Nasal<br>Itching | Sneezing | iTNSS |
|---|---|---|---|---|---|---|---|
| GSP 301 placebo | xx-xxx/xxxxx | Baseline | XX | XX | XX | XX | XX |
| NS pH | | *** | | | | | |
| | | Week 1 | XX | XX | XX | XX | XX |
| | | Week 2 | XX | XX | XX | XX | XX |
| | | Week 3 | XX | XX | XX | XX | XX |
| | | Week 4 | XX | XX | XX | XX | XX |
| | | Week 5 | XX | XX | XX | XX | XX |
| | | Week 6 | XX | XX | XX | XX | XX |
| | | etc | XX | XX | XX | XX | XX |
| | | Week 30 | XX | XX | XX | XX | XX |
| | | etc | XX | XX | XX | XX | XX |
| | | Week 52 | XX | XX | XX | XX | XX |

GSP 301 placebo NS pH GSP 301 NS

iTNSS = sum of four nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing)


Baseline is defined as the average of the last 4 consecutive AM assessments during the last 4 days of the run-in period from the Day -3 AM assessment to the AM assessment on the day of randomization.

Data source: xx

Created on: ddmmmyy hh:mm

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

#### L16.2.6.5 Listing of Change from Baseline of the Average AM Reflective Nasal Symptom Scores (Safety Analysis Set)

| Treatment | Subject /<br>Randomization | | | Nasal | Nasal | | |
|---|---|---|---|---|---|---|---|
| | | Week | Rhinorrhea | | | Ci | -TNICC |
| Group | Number | | Kninorrnea | Congestion | Itching | Sneezing | rTNSS |
| GSP 301 placebo | xx-xxx/xxxxx | Week 1 | XX | XX | XX | XX | XX |
| | | Week 2 | XX | XX | XX | XX | XX |
| | | Week 3 | XX | XX | XX | XX | XX |
| | | Week 4 | XX | XX | XX | XX | XX |
| | | Week 5 | XX | XX | XX | XX | XX |
| | | Week 6 | XX | XX | XX | XX | XX |
| | | etc | XX | XX | XX | XX | XX |
| | | Week 30 | XX | XX | XX | XX | XX |
| | | etc | XX | xx | XX | xx | XX |

GSP 301 placebo NS pH GSP 301 NS

rTNSS = sum of four nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing)

Baseline is defined as the average of the last 4 consecutive AM assessments during the last 4 days of the run-in period from the Day -3 AM assessment to the AM assessment on the day of randomization.

Data source: xx

Created on: ddmmmyy hh:mm


Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### L16.2.6.6 Listing of Change from Baseline of the Average AM Instantaneous Nasal Symptom Scores (Safety Analysis Set)

| Treatment | Subject /<br>Randomization | | | Nasal | Nasal | | |
|---|---|---|---|---|---|---|---|
| Group | Number | Week | Rhinorrhea | Congestion | Itching | Sneezing | iTNSS |
| GSP 301 placebo<br>NS pH | xx-xxx/xxxxx | Week 1 | XX | XX | XX | XX | XX |
| r | | Week 2 | XX | XX | XX | XX | XX |
| | | Week 3 | XX | XX | XX | XX | XX |
| | | Week 4 | XX | XX | XX | XX | XX |
| | | Week 5 | XX | XX | XX | XX | XX |
| | | Week 6 | XX | XX | XX | XX | XX |
| | | etc | XX | XX | XX | XX | XX |
| | | Week 30 | XX | XX | XX | XX | XX |
| | | etc | xx | xx | XX | xx | XX |

GSP 301 placebo NS pH GSP 301 NS

iTNSS = sum of four nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing)

Baseline is defined as the average of the last 4 consecutive AM assessments during the last 4 days of the run-in period from the Day -3 AM assessment to the AM assessment on the day of randomization.

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

|---|---|
| (Study No. GSP 301-303) | r |

# L16.2.6.7 Listing of Rhinoconjunctivitis Quality of Life (RQLQ(S)) (Part I) (Safety Analysis Set)

| Treatment<br>Group | Subject / | | ActivitiesSleep | | | | | Non-Nose/EyeSymptom | | | | | | Practical Problem | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Randomization<br>Number | Visit | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q7 | Q8 | Q9 | Q10 | Q11 | Q12 | Q13 | Q14 | Q15 | Q16 |
| GSP 301 placebo<br>NS pH | xx-xxx/xxxxx | Visit 2 | Х | X | X | X | X | X | X | X | X | Х | X | Х | X | Х | Х | X |
| 1 | | Visit 4 | X | X | X | X | X | X | X | X | X | X | X | X | X | x | X | X |
| | | Visit 8 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| | | Visit<br>12 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

GSP 301 placebo NS pH GSP 301 NS

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# $L16.2.6.7 \ Listing \ of \ Rhinoconjunctivitis \ Quality \ of \ Life \ (RQLQ(S)) \ (Part \ II)$ $(Safety \ Analysis \ Set)$

| T | Subject / | | Nasal Symptom | | | Eye<br>Symptom | | | Emotional | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Randomization<br>Number | Visit | Q17 | Q18 | Q19 | Q20 | Q21 | Q22 | Q23 | Q24 | Q25 | Q26 | Q27 | Q28 |
| GSP 301 placebo | xx-xxx/xxxxx | Visit 2 | Х | Х | Х | Х | Х | х | х | X | Х | х | Х | X |
| | | Visit 4 | X | x | x | X | X | X | X | X | x | X | X | X |
| | | Visit 8 | X | X | X | X | X | X | X | X | X | X | X | X |
| | | Visit<br>12 | X | X | X | X | X | X | X | X | X | X | X | X |

GSP 301 placebo NS pH GSP 301 NS

Data source: xx

Glenmark 

|---|---|---|

#### L16.2.6.8 Listing of Rhinoconjunctivitis Quality of Life (RQLQ(S)) by Domain (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Visit | Activities | Sleep | Non-<br>Nose/Eye<br>Symptom | Practical<br>Problem | Nasal<br>Symptom | Eye<br>Symptom | Emotional | Overall<br>Average<br>RQLQ |
|---|---|---|---|---|---|---|---|---|---|---|
| GSP 301 placebo | xx-xxx/xxxxx | Visit 2 | XX | XX | xx | xx | xx | XX | XX | XX |
| 1 | | Visit 4 | XX | XX | XX | XX | XX | XX | XX | XX |
| | | Visit 8 | XX | XX | XX | XX | XX | XX | XX | XX |
| | | Visit 12 | XX | XX | XX | XX | XX | XX | XX | XX |

GSP 301 placebo NS pH GSP 301 NS

A domain average score is calculated as the sum of the scores in that domain divided by the number of items in that domain.

The overall average RQLQ(S) score is calculated as the sum of the scores in all domains divided by the total number of items in the seven domains.

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

#### $L16.2.6.9 \ Listing \ of \ Change \ from \ Baseline \ in \ Rhinoconjunctivitis \ Quality \ of \ Life \ (RQLQ(S)) \ by \ Domain \ (Safety \ Analysis \ Set)$

| | Subject / | | | | Non- | | | | | Overall |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Randomization | | | | Nose/Eye | Practical | Nasal | Eye | | Average |
| Group | Number | Visit | Activities | Sleep | Symptom | Problem | Symptom | Symptom | Emotional | RQLQ |
| GSP 301 placebo | xx-xxx/xxxxx | Visit 4 | XX | XX | XX | XX | XX | XX | XX | XX |
| NS pH | | | | | | | | | | |
| | | Visit 8 | XX | XX | XX | XX | XX | XX | XX | XX |
| | | Visit 12 | XX | XX | XX | XX | XX | XX | XX | XX |

GSP 301 placebo NS pH GSP 301 NS

Baseline is defined as the RQLQ(S) score at the Randomization Visit (Visit 2).

A domain average score is calculated as the sum of the scores in that domain divided by the number of items in that domain.

The overall average RQLQ(S) score is calculated as the sum of the scores in all domains divided by the total number of items in the seven domains.

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
| (Study No. GSP 301-303) | | |

# L16.2.6.10 Listing of Physician Assessed Nasal Symptom Scores (PNSS) (Safety Analysis Set)

| | Subject / | | | | | | |
|---|---|---|---|---|---|---|---|
| Treatment | Randomization | | | Nasal | Nasal | | |
| Group | Number | Visit | Rhinorrhea | Congestion | Itching | Sneezing | PNSS |
| GSP 301 placebo NS pH | xx-xxx/xxxxx | Visit 2 | 0 | 1 | 1 | 0 | 2 |
| | | Visit 3 | 0 | 0 | 1 | 0 | 1 |
| | | Visit 4 | 0 | 1 | 0 | 0 | 1 |
| | | etc | 0 | 0 | 0 | 0 | 0 |

GSP 301 placebo NS pH GSP 301 NS

PNSS = sum of four nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing)

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

### L16.2.6.11 Listing of Change from Baseline in Physician Assessed Nasal Symptom Scores (PNSS) (Safety Analysis Set)

| Treatment | Subject /<br>Randomization | | | Nasal | Nasal | | |
|---|---|---|---|---|---|---|---|
| Group | Number | Visit | Rhinorrhea | Congestion | Itching | Sneezing | PNSS |
| GSP 301 placebo NS pH | xx-xxx/xxxxx | Visit 3 | XX | XX | xx | xx | XX |
| - • | | etc | XX | XX | XX | XX | XX |

GSP 301 placebo NS pH GSP 301 NS

PNSS = sum of four nasal symptom scores (Rhinorrhea, Nasal Congestion, Nasal Itching, Sneezing) Baseline is defined as the symptom score at the Randomization Visit (Visit 2).

Data source: xx

 $\label{eq:created on: ddmmmyy hh:mm} Page \ 1 \ of \ N$ 

Glenmark 

|---|---|
| (Study No. GSP 301-303) | r |

#### L16.2.6.12 Listing of Rhinitis Control Assessment Test (RCAT) (Safety Analysis Set)

| Treatment | Subject /<br>Randomization | | Domain | Domain | Domain | Domain | Domain | Domain | Total |
|---|---|---|---|---|---|---|---|---|---|
| Group | Number | Visit | 1 | 2 | 3 | 4 | 5 | 6 | RCAT |
| GSP 301 placebo NS pH | xx-xxx/xxxxx | Visit 2 | 0 | 1 | 1 | 0 | 2 | 2 | 6 |
| • | | Visit 4 | 0 | 0 | 1 | 0 | 1 | 2 | 4 |
| | | Visit 8 | 0 | 1 | 0 | 0 | 0 | 0 | 1 |
| | | Visit 12 | 0 | 0 | 0 | 0 | 2 | 0 | 2 |

GSP 301 placebo NS pH GSP 301 NS

Total RCAT score is calculated by adding individual scores for each RCAT item. The total RCAT score can range from 6 to 30.

Data source: xx

Created on: ddmmmyy hh:mm  $Page \ 1 \ of \ N$ 

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

#### L16.2.6.13 Listing of Change from Baseline in Rhinitis Control Assessment Test (RCAT) (Safety Analysis Set)

| Treatment | Subject /<br>Randomization | | Domain | Domain | Domain | Domain | Domain | Domain | Total |
|---|---|---|---|---|---|---|---|---|---|
| Group | Number | Visit | 1 | 2 | 3 | 4 | 5 | 6 | RCAT |
| GSP 301 placebo NS | xx-xxx/xxxxx | Visit 4 | 0 | -1 | 0 | 0 | -1 | 0 | -2 |
| рН | | Visit 8 | 0 | 0 | -1 | 0 | -2 | -2 | -5 |
| 1 | | Visit 12 | 0 | -1 | -1 | 0 | 0 | -2 | -4 |

GSP 301 placebo NS pH GSP 301 NS

Total RCAT score is calculated by adding individual scores for each RCAT item. The total RCAT score can range from 6 to 30. Baseline is defined as the domain score at the Randomization Visit (Visit 2).

Data source: xx

Glenmark 

|---|---|
| (Study No. GSP 301-303) | r |

# L16.2.7.1 Listing of Treatment Emergent Adverse Events by Treatment During Randomized Treatment Period (Safety Analysis Set)

#### GSP 301 placebo NS pH

| Subject /<br>Randomization<br>Number | AE<br>No. | Body System/<br>MedDRA Term/<br>AE Term | Start /End<br>Date | Severity | Relationship<br>to Study<br>Medication | Outcome | Action<br>Taken<br>with IP | Other<br>Action<br>Taken | Serious<br>AE? |
|---|---|---|---|---|---|---|---|---|---|
| xx-xxx/xxxxx | XX | NERVOUS SYSTEM<br>DISORDERS/ HEADACHE/<br>HEADACHE | 2012-10-12/<br>2012-10-15 | Mild | Not Related | Improved | None | None | No |

Programming note: table will continue for GSP 301 placebo NS pH and GSP 301 NS

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

#### L16.2.7.2 Listing of Adverse Events During Placebo Run-in Period

| Subject /<br>Randomization<br>Number | AE<br>No. | Body System/<br>MedDRA Term/<br>AE Term | Start /End<br>Date | Severity | Relationship<br>to Study<br>Medication | Outcome | Action<br>Taken<br>with IP | Other<br>Action<br>Taken | Serious<br>AE? |
|---|---|---|---|---|---|---|---|---|---|
| xx-xxx/xxxxx | XX | NERVOUS SYSTEM<br>DISORDERS/ HEADACHE/<br>HEADACHE | 2012-10-12/<br>2012-10-15 | Mild | Not Related | Recovered/Res<br>olved | None | None | No |

Data source: xx

Created on: ddmmmyy hh:mm


Glenmark 

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 011pt 2017 |

# L16.2.7.3 Listing of Pre-Treatment Adverse Events (Safety Analysis Set)

| Subject / | | Body System/ | | | Relationship | | Action | Other | Serious |
|---|---|---|---|---|---|---|---|---|---|
| Randomization | AΕ | MedDRA Term/ | Start /End | | to Study | | Taken | Action | AE? |
| Number | No. | AE Term | Date | Severity | Medication | Outcome | with IP | Taken | |
| xx-xxx/xxxxx | XX | NERVOUS SYSTEM<br>DISORDERS/ HEADACHE/ | 2012-10-12/<br>2012-10-15 | Mild | Not Related | Improved | None | None | No |
| | | HEADACHE | | | | | | | |

Data source: xx

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# L16.2.8.1 Listing of Clinical Laboratory Test Results (Biochemistry) (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Visit | Date /Time | Lab<br>Test | Results | Unit | Normal<br>Range | Flag/<br>Significance<br>(CS/NCS) |
|---|---|---|---|---|---|---|---|---|
| GSP 301 placebo<br>NS pH | xx-xxx/xxxxx | Visit 1 | ddmmmyyy h:mm | ALBUMIN | 46 | g/L | 30 - 50 | Normal |
| NS рн | | *** | | BILIRUBIN<br>etc | 1.6 | mg/dL | 0.2 - 1.2 | High (NCS) |

Visit 8 Visit 12

GSP 301 placebo NS pH GSP 301 NS

CS= Clinically Significant; NCS= Not Clinically Significant;

Data source: xx Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 011pt 2017 |

# L16.2.8.2 Listing of Clinical Laboratory Test Results (Hematology) (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Visit | Date /Time | Lab<br>Test | Results | Unit | Normal<br>Range | Flag/<br>Significance<br>(CS/NCS) |
|---|---|---|---|---|---|---|---|---|
| GSP 301 placebo | xx-xxx/xxxxx | Visit 1 | ddmmmyyy h:mm | RBC | XXX | XXX | xx - xxx | Normal |
| NS pH | | Visit 8<br>Visit 12 | | WBC<br>etc | XXX | xxx | XX - XXX | Normal |
| GSP 301 placebo NS pH<br>GSP 301 NS | | | | | | | | |

CS= Clinically Significant; NCS= Not Clinically Significant;

Data source: xx Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# L16.2.8.3 Listing of Clinical Laboratory Test Results (Urinalysis) (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Visit | Date /Time | Lab<br>Test | Results | Unit | Normal<br>Range | Flag/<br>Significance<br>(CS/NCS) |
|---|---|---|---|---|---|---|---|---|
| GSP 301 placebo | xx-xxx/xxxxx | Visit 1 | ddmmmyyy h:mm | XXX | XXX | XXX | xx - xxx | Normal |
| NS pH | | | | | | | | |
| • | | | | XXX | XXX | XXX | xx - xxx | Normal |
| | | | | etc | | | | |
| | | Visit 8 | | | | | | |
| | | Visit 12 | | | | | | |

GSP 301 placebo NS pH GSP 301 NS

CS= Clinically Significant; NCS= Not Clinically Significant;

Data source: xx Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 011pt 2017 |

# L16.2.8.4 Listing of Pregnancy Test Results (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Visit | Date | Result | Reason Not done |
|---|---|---|---|---|---|
| GSP 301 placebo NS pH | xx-xxx/xxxxx | Visit 1<br>Visit 2<br>Visit 3 | ddmmmyyyy | Negative<br>Negative | xxxxxxxxxxxxxx |
| | | Visit 4<br>etc<br>Visit 12 | ddiiiiiiiyyyy | Negative | |
| GSP 301 placebo NS pH<br>GSP 301 NS | | | | | |

Data source: xx Created on: ddmmmyy hh:mm


Glenmark 

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 011pt 2017 |

# L16.2.8.5 Listing of Vital Signs (Safety Analysis Set)

| Treatment | Subject /<br>Randomization<br>Number | Visit | Test | Rogult | Unit | Normal/<br>Abnormal<br>(CS/NCS) |
|---|---|---|---|---|---|---|
| GCD 201 rds adv NG rd | | Visit1 | | Result<br>126/70 | mmHg | |
| GSP 301 placebo NS pH | xx-xxx/xxxxx | Visit 2 Visit 8 Visit 12 | Blood Pressure (Sitting) Pulse Rate Body Weight Height Blood Pressure (Sitting) Pulse Rate | 118<br>62.5<br>168<br>xxx/xxx<br>xxx | bpm<br>kg<br>cm<br>mmHg<br>bpm | Normal<br>Abnormal (NCS) |
| GSP 301 placebo NS pH<br>GSP 301 NS | | | | | | |

CS= Clinically Significant; NCS= Not Clinically Significant;

Data source: xx Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

| | rsion Number: | SAP Version Date: |
|---|---|---|
| GPL/CT/2014/018/III Version (Study No. GSP 301-303) | 1.0 | 04-Apr-2017 |

# L16.2.8.6 Listing of 12-Lead ECGs (Safety Analysis Set)

| | andomization<br>umber | Visit | Date | Rate (bpm) | Interval<br>(ms) | Interval<br>(ms) | Duration<br>(ms) | Interval<br>(ms) | Interval<br>(ms) | Abnormal<br>(CS/NCS) |
|---|---|---|---|---|---|---|---|---|---|---|
| GSP 301 placebo xx<br>NS pH | | | ddmmmyyy | xxx | xxx<br>xxx | xxx | xxx | xxx | xxx<br>xxx | Normal Abnormal (NCS) |

GSP 301 placebo NS pH GSP 301 NS

CS= Clinically Significant; NCS= Not Clinically Significant;

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

# L16.2.8.7 Listing of Physical Examination (Safety Analysis Set)

| Treatment | Subject /<br>Randomization | | | Normal/<br>Abnormal | |
|---|---|---|---|---|---|
| Group | Number | Visit | Body System | (CS/NCS) | Comments |
| GSP 301 placebo NS pH | XX-XXX/XXXXX | Visit 1 Visit 8 Visit 12 | General Appearance Neck Head and Eyes Cardiovascular Lungs and Thorax Abdominal and Gastro-Enteric Neurological Dermatological Musculoskeletal and Extremities | Normal<br>Normal<br>Abnormal (NCS)<br>Normal<br>Normal<br>Normal | |
| GSP 301 placebo NS pH<br>GSP 301 NS | | | | | |

CS= Clinically Significant; NCS= Not Clinically Significant;

Data source: xx

Created on: ddmmmyy hh:mm  $\qquad \qquad \text{Page 1 of N}$ 

Glenmark 

|---|---|
| (Study No. GSP 301-303) | r |

# L16.2.8.8 Listing of Focused ENT Examination (Safety Analysis Set)

| Treatment Grading (Scale) or Significan Group Number Visit Evaluation Results (CS/NCS) GSP 301 placebo NS pH Xx-xxx/xxxx | | Randomization | | | Grading (Scale) or | |
|---|---|---|---|---|---|---|
| GSP 301 placebo NS pH xx-xxx/xxxxx Visit 1 Nasal Irritation Epistaxis 1 (Mild) Mucosal Edema 1 (Mild) Mucosal Erythema Crusting Of Mucosa 0 (None) Nasal Discharge Throat Irritation Candidiasis Post Nasal Drip Visit 2 etc 1 (Mild) O (None) (None) (None) (None) (Absent) (Absent) | Cuara | | | | | |
| Epistaxis 1 (Mild) Mucosal Edema 1 (Mild) Mucosal Erythema 0 (None) Crusting Of Mucosa 0 (None) Nasal Discharge 0 (None) Throat Irritation 0 (Absent) Candidiasis 0 (Absent) Post Nasal Drip 0 (Absent) Visit 2 etc | Group | Number | Visit | Evaluation | Results | (CS/NCS) |
| Mucosal Edema 1 (Mild) Mucosal Erythema 0 (None) Crusting Of Mucosa 0 (None) Nasal Discharge 0 (None) Throat Irritation 0 (Absent) Candidiasis 0 (Absent) Post Nasal Drip 0 (Absent) Visit 2 etc | GSP 301 placebo NS pH | xx-xxx/xxxxx | Visit 1 | Nasal Irritation | 1B (Superficial mucosal erosion) | |
| Mucosal Erythema 0 (None) Crusting Of Mucosa 0 (None) Nasal Discharge 0 (None) Throat Irritation 0 (Absent) Candidiasis 0 (Absent) Post Nasal Drip 0 (Absent) Visit 2 etc | · · · | | | Epistaxis | 1 (Mild) | |
| Crusting Of Mucosa 0 (None) Nasal Discharge 0 (None) Throat Irritation 0 (Absent) Candidiasis 0 (Absent) Post Nasal Drip 0 (Absent) Visit 2 etc | | | | Mucosal Edema | 1 (Mild) | |
| Nasal Discharge 0 (None) Throat Irritation 0 (Absent) Candidiasis 0 (Absent) Post Nasal Drip 0 (Absent) Visit 2 etc | | | | Mucosal Erythema | 0 (None) | |
| Throat Irritation 0 (Absent) Candidiasis 0 (Absent) Post Nasal Drip 0 (Absent) Visit 2 etc | | | | Crusting Of Mucosa | 0 (None) | |
| Candidiasis 0 (Absent) Post Nasal Drip 0 (Absent) Visit 2 etc | | | | Nasal Discharge | 0 (None) | |
| Post Nasal Drip 0 (Absent) Visit 2 etc | | | | Throat Irritation | 0 (Absent) | |
| Visit 2 etc | | | | Candidiasis | 0 (Absent) | |
| etc | | | | Post Nasal Drip | 0 (Absent) | |
| | | | Visit 2 | | | |
| Visit 12 | | | etc | | | |
| | | | Visit 12 | | | |

GSP 301 NS

CS= Clinically Significant; NCS= Not Clinically Significant;

Data source: xx Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

|---|---|
| (Study No. GSP 301-303) | r |

# L16.2.8.9 Listing of Eye Examination (Safety Analysis Set)

| Treatment<br>Group | Subject /<br>Randomization<br>Number | Visit | Eye Examination<br>Date | Results<br>Right Eye | Results<br>Left Eye |
|---|---|---|---|---|---|
| GSP 301 placebo NS pH | xx-xxx/xxxxx | Visit 1<br>Visit 2<br>Visit 3<br>Visit 4<br>etc<br>Visit 12 | ddmmmyyyy | Normal | Normal |
| GSP 301 placebo NS pH<br>GSP 301 NS | | | | | |

Data source: xx

Created on: ddmmmyy hh:mm Page 1 of N

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III | X7 ' 1.0 | SAP Version Date: |
|-----------------------------------------|--------------|-------------------|
| (Study No. GSP 301-303) | V CISION 1.0 | 04-Apr-2017 |

F15.1.1 LS Means with 95% CIs of of AM Average rTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)



Programming note: For the LS means plots, please maintain consistency over y-axis range for endpoints. For example for TNSS outputs, ensure the y-axis range is the same in case various outputs need comparing.

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
| (Study No. GSP 301-303) | | |

#### F15.1.2 LS Means with 95% CIs of of AM Average rTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set) Repeat of F15.1.1 for Per Protocol Set

#### F15.1.3 LS Means with 95% CIs of of AM Average iTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)

Repeat of F15.1.1 for iTNSS Full Analysis Set

F15.1.4 LS Means with 95% CIs of of AM Average iTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set)

Repeat of F15.1.1 for iTNSS Per Protocol Set

 $F15.1.5\;LS$  Means with 95% CIs of Overall RQLQ(S) at Weeks 6, 30, and 52 (Full Analysis Set)

Repeat of F15.1.1 for RQLQ(S) Full Analysis Set

Glenmark 

|-------------------------|-------------------|
| (Study No. GSP 301-303) | 0171pi 2017 |

F15.2.1 Treatment Differences of LS Means with 95% CIs of AM Average rTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)



Programming note: For the treatment differences of LS means plots, please maintain consistency over y-axis range for endpoints. For example for TNSS outputs, ensure the y-axis range is the same in case various outputs need comparing.

Glenmark 

|---|---|
| (Study No. GSP 301-303) | r |

F15.2.2 Treatment Differences of LS Means with 95% CIs of AM Average rTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set)

Repeat of F15.2.1 for Per Protocol Set

F15.2.3 Treatment Differences of LS Means with 95% CIs of AM Average iTNSS over the First 6, 30, and 52 Weeks of Treatment (Full Analysis Set)
Repeat of F15.2.1 for iTNSS Full Analysis Set

F15.2.4 Treatment Differences of LS Means with 95% CIs of AM Average iTNSS over the First 6, 30, and 52 Weeks of Treatment (Per Protocol Set)

Repeat of F15.2.1 for iTNSS Per Protocol Set

F15.2.5 Treatment Differences of LS Means with 95% CIs of Overall RQLQ(S) at Weeks 6, 30, and 52 (Full Analysis Set)
Repeat of F15.2.1 for RQLQ(S) Full Analysis Set

Glenmark 

| Protocol Number:<br>GPL/CT/2014/018/III<br>(Study No. GSP 301-303) | SAP Version Number:<br>Version 1.0 | SAP Version Date:<br>04-Apr-2017 |
|---|---|---|
|---|---|---|

F15.3.1 LS Means with 95% CIs of Average AM rTNSS over each Treatment Week (Full Analysis Set)



Programming note: An offset will be applied to the treatments to prevent an overlap of treatment information. Offset values TBD during programming'. An example at the time of programming could be the following: GSP 301 could have an offset of -0.1 and placebo of +0.1, so to plot the treatment information at week 28, the x-value for GSP 301 will be 27.9 and placebo will be 28.1, but again a visual check needs to be applied to see how practical/appropriate the plot looks.

F15.3.2 LS Means with 95% CIs of Average AM iTNSS over each Treatment Week (Full Analysis Set)

Repeat of F15.3.1 for iTNSS

Glenmark 

|-------------------------|-------------------|
| (Study No. GSP 301-303) | r |

F15.4.1 Treatment Differences of LS Means with 95% CIs of AM Average rTNSS over each Treatment Week (Full Analysis Set)



F15.4.2 Treatment Differences of LS Means with 95% CIs of AM Average iTNSS over each Treatment Week (Full Analysis Set)

Repeat of F15.4.1 for iTNSS

Glenmark 




04-Apr-2017

#### **Reference:**

1. Center for Drug Evaluation and Research. Guidance for Industry. Allergic Rhinitis: Clinical Development Programs for Drug Products. Apr 2000.




04-Apr-2017

#### Appendix 2

#### **Schedule of Procedures and Assessments**

| Visits | Screen | Randomiz | | | Τ | reatm | ent Vi | sits (T | V) | | | Final Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | ing | ation Visit | TV | TV | TV | TV | TV | TV | TV | TV | TV | / |
| | Visit | (RV) | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | Discontinu |
| | (SV) | Visit 2 | | | | | | | | | | ation |
| | Visit 1 | | | | | | | | | | | Visit |
| | | | | | | | | | | | | (FV/DV) |
| | | | | | | | | | | | | Visit 12 |
| Week | -1 | 1 | 3 | 6 | 12 | 18 | 24 | 30 | 36 | 42 | 48 | 52 |
| Day ± Window | (-7 to - | 1 | 22± | 43± | 85± | 127 | 169 | 211 | 253 | 295 | 337 | 365+10 |
| | 10) | | 3 | 3 | 5 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | |
| Activity / Observation | | | | | | | | | | | | |
| Written informed consent | X | | | | | | | | | | | |
| (assent, if applicable) and | | | | | | | | | | | | |
| HIPAA authorization | | | | | | | | | | | | |
| Inclusion/exclusion | X | | | | | | | | | | | |
| criteria review | | | | | | | | | | | | |
| Demographic data | X | | | | | | | | | | | |
| Medical & treatment | X | | | | | | | | | | | |
| history | | | | | | | | | | | | |
| Concomitant medication | X | X | X | X | X | X | X | X | X | X | X | X |
| evaluation | | | | | | | | | | | | |
| Physical examination | X | | | | | | | X | | | | X |
| Vital signs | X | X | | | | | | X | | | | X |
| Height and weight | X | | | | | | | X | | | | X |
| measurements | | | | | | | | | | | | |
| Clinical laboratory | X | | | | | | | X | | | | X |
| investigations | | | | | | | | | | | | |
| (hematology, | | | | | | | | | | | | |
| biochemistry, urinalysis) <sup>a</sup> | | | | | | | | | | | | |
| Focused ENT and eye | X | X | X | X | X | X | X | X | X | X | X | X |
| examination <sup>b</sup> | | | | | | | | | | | | |
| Allergen testing (skin | X | | | | | | | | | | | |
| prick test for relevant | | | | | | | | | | | | |
| allergen, if required) <sup>c</sup> | | | | | | | | | | | | |
| 12-lead ECG | X | | | | | | | | | | | X |
| Urine pregnancy test (if | X | X | X | X | X | X | X | X | X | X | X | X |
| applicable) | | | | | | | | | | | | |



Protocol Number: GPL/CT/2014/018/III (Study No. GSP 301-303) SAP Version Number: SAP Version Date: Version 1.0

04-Apr-2017

| Visits | Screen | Randomiz | | | T | reatm | ent Vis | sits (TV | V) | | | Final Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | ing<br>Visit<br>(SV)<br>Visit 1 | ation Visit<br>(RV)<br>Visit 2 | TV<br>3 | TV<br>4 | TV<br>5 | TV 6 | TV 7 | TV<br>8 | TV<br>9 | TV<br>10 | TV<br>11 | Discontinu ation Visit (FV/DV) |
| Week | -1 | 1 | 3 | 6 | 12 | 18 | 24 | 30 | 36 | 42 | 48 | Visit 12<br>52 |
| Day ± Window | (-7 to -<br>10) | 1 | 22±<br>3 | 43±<br>3 | 85±<br>5 | 127<br>±7 | 169<br>±7 | 211<br>±7 | 253<br>±7 | 295<br>±7 | 337<br>±7 | 365+10 |
| Review instructions and train on the proper use of the nasal spray using the GSP 301 placebo NS pH bottle | X | | | | | | | | | | | |
| Review instructions and train on the proper use of the nasal spray | | X | X | X | X | X | X | X | X | X | X | |
| Prime and dispensation<br>and administration of<br>single-blind GSP 301<br>placebo NS pH at the<br>clinic <sup>d</sup> | X | | | | | | | | | | | |
| Return single-blind GSP 301 placebo NS pH to the clinic <sup>e</sup> | | X | | | | | | | | | | |
| Distribution of the AR Assessment Diary | X | X | X | X | X | X | X | X | X | X | X | |
| Collection/Review of the AR Assessment Diary | | X | X | X | X | X | X | X | X | X | X | X |
| Subject assessment of AR symptoms and recording and self-administration of placebo run-in medication <sup>d</sup> | X <sup>d</sup> _ | <del></del> | | | | | | | | | | |
| Subject assessment of AR symptoms and recording and self-administration of double-blind study medication <sup>d</sup> | | х | | | | | | | | | | <b>→</b> |
| Physician assessment of nasal symptom severity | | X | X | X | X | X | X | X | X | X | X | X |
| Review randomization criteria | | X | | | | | | | | | | |

| AD-D51-05.02 25-Jan-2015 Confidential Fage 150 01 152 | AD-BST-05.02 23-Jan-2015 | Confidential |
|---|---|---|
|---|---|---|




X

X

X

X

X

X

X

Protocol Number: GPL/CT/2014/018/III (Study No. GSP 301-303)

RQLQ(S)<sup>f</sup> RCAT

Adverse

monitoring

Subject compliance check

SAP Version Number:

04-Apr-2017


Visits Screen Randomiz **Treatment Visits (TV) Final Visit** ing ation Visit TVTVTVTVTVTVTV TVTV5 7 10 Discontinu Visit (RV) 3 4 6 8 9 11 Visit 2 (SV) ation Visit 1 Visit (FV/DV) Visit 12 Week 3 12 18 24 30 36 42 48 52 -1 1 6 Day ± Window (-7 to -1 253 295 22± 43±  $85\pm$ 127 169 211 337 365+10 ±7 10) 3 5 ±7 ±7 ±7 ±7 ±7 3 X Randomization/treatment assignment Χ Χ Prime and dispensation of Χ X X X X X X X double-blind study medication Administration of double-X blind study medication at the clinic<sup>d</sup> X Return double-blind study X X X X X X X X X medication to the clinic<sup>e</sup> Distribution of X X X X the RQLQ(S), review instructions with the subject, and subject completion of the

Abbreviations: AM = morning; AR = allergic rhinitis; ECG = electrocardiogram; ENT = ears, nose, and throat; HIPAA = Health Insurance Portability and Accountability Act; NS = nasal spray; RQLQ(S) = Rhinoconjunctivitis Quality of Life Questionnaire - Standardized Activities; RCAT = Rhinitis Control Assessment Test.

X

X

X

X

X

X

Χ

a: Refer to Appendix 3 for the list of clinical laboratory tests.

X

events

X

X

b: A focused ENT and eye examination will be done at all visits. Focused nasal examinations will be performed to assess signs of AR as well as known complications of intranasal corticosteroid or antihistamine use (i.e., bleeding, perforation, and ulceration). Throat examinations will be conducted to evaluate evidence of throat irritation and candidiasis. If at any visit, clinically significant nasal ulceration, nasal mucosal erosion, and nasal septal perforation are observed, or a finding at a previous visit has worsened (as judged by the Investigator), the subject should be referred to a qualified ENT specialist or other medically qualified specialist (qualified to evaluate and record these conditions, as judged by the Investigator) for further evaluation. A record from the specialist should be maintained, including the photographic evidence (imaging of nasal mucosa) of the assessment to allow pre- and post-treatment comparisons for AEs. The Sponsor will collect the de-identified information as part of the study data collection. Eligibility of the subject for participation/continued participation in the study will be at the Investigator's discretion based on whether or not the protocol-defined selection criteria are met. These subjects may need to be re-screened due to delay in scheduling an ENT visit to obtain the necessary evaluation, as applicable, upon consultation with

| AD-BST-05.02 23-Jan-2015 Confidential Page 151 of |
|---------------------------------------------------|
|---------------------------------------------------|



Protocol Number: GPL/CT/2014/018/III (Study No. GSP 301-303) SAP Version Number: SAP Version Date: Version 1.0 04-Apr-2017

the Sponsor's study team and approval. A thorough eye examination will also be performed by the Investigator or medically qualified designee to assess signs of AR as well as any known complications of intranasal corticosteroid or antihistamine use. If needed, the subject should be referred to a qualified ophthalmologist for further evaluation as soon as possible.

- c: Documentation of a positive result within the last year (12 months) before the Screening Visit (Visit 1) is acceptable to meet the eligibility criteria. Intradermal and/or RAST testing will not be accepted.
- d: Generally, subjects will assess/record AR symptoms and take study medication at home. Subjects will assess their symptoms at specified clinic visits, as directed by the site personnel. The subject assessment and recording of AR symptoms will be done at the clinic at the Screening Visit (Visit 1) and study medication will be self-administered in the clinic at the Screening Visit (Visit 1) and the Randomization Visit (Visit 2) doses of study medication during the run-in and treatment periods should be taken immediately following completion of the AR Assessment Diary (as applicable) except on the morning of the Screening Visit (Visit 1) and Randomization Visit (Visit 2) when the first dose of the placebo run-in medication and the double-blind study medication, respectively, will be self-administered in the clinic under the supervision of site personnel. doses of study medication should be taken approximately At the Screening Visit (Visit 1), subjects should be told not to take study medication before com ng to the clinic for the Randomization Visit (Visit 2). The last dose of the double-blind study medication should be the lose on the day before the Final Visit/Discontinuation Visit (Visit 12). Subjects should be reminded not to take study medication on the morning of the Final Visit/Discontinuation Visit (Visit 12).
- e: Subjects should be instructed to bring their study medication kit to each visit after the Screening Visit (Visit 1). Site personnel will collect the kit, take the used study medication, and return the rest of the kit to the subject, as applicable. f: The RQLQ(S) must be the first procedure conducted at these visits.